CLINICAL TRIAL: NCT05000216
Title: Booster Effects With Autoimmune Treatments in Patients With Poor Response to Initial COVID-19 Vaccine (ACV01)
Brief Title: COVID-19 Booster Vaccine in Autoimmune Disease Non-Responders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed due to continued enrollment hurdles.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAIT ACV01; NIAID CRMS ID#: 38873 (Other: DAIT NIAID)
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA); Systemic Lupus Erythematosus (SLE); Pemphigus Vulgaris; Multiple Sclerosis (MS); Systemic Sclerosis (SSc); Pediatric SLE; Juvenile Idiopathic Arthritis (JIA); Juvenile Dermatomyositis (JDM); Pediatric-Onset Multiple Sclerosis (POMS)
Keywords: SARS-CoV-2 Infection; COVID-19; autoimmune disease; non-responders to COVID-19 vaccination; suboptimal response to COVID-19 vaccination; COVID-19 booster vaccine; booster effects with autoimmune treatments
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Pemphigus; Multiple Sclerosis; Scleroderma, Systemic; Arthritis, Juvenile; Dermatomyositis; COVID-19; Autoimmune Diseases | interventions — 2019-nCoV Vaccine mRNA-1273; COVID-19 Vaccines; BNT162 Vaccine; Ad26COVS1; Mycophenolic Acid; Methotrexate; BNT162b5

STUDY DESIGN:
Intervention Model Description: Adults and Pediatrics
  Stage 1: Participants in Cohorts A and B will be randomized into two immunosuppressive (IS) medication treatment plans as follows:
  * Participants continue to take their cohort-defining IS medications without alterations in schedule and dosing
  * Participants withhold their cohort-defining IS medications before and after additional homologous vaccine dose, per protocol instruction
  * Cohort C: No randomization-Participants continue to take their IS medications without alterations in schedule and dosing.
    * Stage 2: Participants in Cohorts D and E will withhold their cohort-defining IS medications before and after additional alternative vaccine dose, per protocol instruction. Cohort F: No randomization-Participants withhold their IS medications before and after additional alternative vaccine dose, per protocol instruction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (43):
- Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) (Experimental): Adult participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will receive an additional dose of the Moderna COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Moderna mRNA-1273; Drug: Continue IS (MMF or MPA)
- Cohort A, Arm A2: BNT162b2 + Continue IS (MMF or MPA) (Experimental): Adult participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will receive an additional dose of the Pfizer-BioNTech COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: BNT162b2; Drug: Continue IS (MMF or MPA)
- Cohort A, Arm A3: Ad26.COV2.S + Continue IS (MMF or MPA) (Experimental): Arm closed, effective protocol version 3.0. Adult participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will receive the Janssen COVID-19 vaccine booster (1 dose) and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Ad26.COV2.S; Drug: Continue IS (MMF or MPA)
- Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) (Experimental): Adult participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Moderna mRNA-1273; Drug: Withhold IS (MMF or MPA)
- Cohort A, Arm A5: BNT162b2 + Withhold IS (MMF or MPA) (Experimental): Adult participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Pfizer-BioNTech COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: BNT162b2; Drug: Withhold IS (MMF or MPA)
- Cohort A, Arm A6: Ad26.COV2.S + Withhold IS (MMF or MPA) (Experimental): Arm closed, effective protocol version 3.0. Adult participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after the Janssen COVID-19 vaccine booster (1 dose), per protocol instruction.
  Interventions: Biological: Ad26.COV2.S; Drug: Withhold IS (MMF or MPA)
- Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) (Experimental): Adult participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will receive an additional dose of the Moderna COVID-19 vaccine booster and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Moderna mRNA-1273; Drug: Continue IS (MTX)
- Cohort B, Arm B2: BNT162b2 + Continue IS (MTX) (Experimental): Adult participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will receive an additional dose of the Pfizer-BioNTech COVID-19 vaccine booster and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: BNT162b2; Drug: Continue IS (MTX)
- Cohort B, Arm B3: Ad26.COV2.S + Continue IS (MTX) (Experimental): Arm closed, effective protocol version 3.0. Adult participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will receive the Janssen COVID-19 vaccine booster (1 dose) and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Ad26.COV2.S; Drug: Continue IS (MTX)
- Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) (Experimental): Adult Participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Moderna mRNA-1273; Drug: Withhold IS (MTX)
- Cohort B, Arm B5: BNT162b2 + Withhold IS (MTX) (Experimental): Adult participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Pfizer-BioNTech COVID-19 vaccine booster, per protocol instruction.
  Interventions: Biological: BNT162b2; Drug: Withhold IS (MTX)
- Cohort B, Arm B6: Ad26.COV2.S + Withhold IS (MTX) (Experimental): Arm closed, effective protocol version 3.0. Adult participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after the Janssen COVID-19 vaccine booster (1 dose), per protocol instruction.
  Interventions: Biological: Ad26.COV2.S; Drug: Withhold IS (MTX)
- Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (B cell depletion therapy) (Experimental): Adult participants taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will receive an additional dose of the Moderna COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Moderna mRNA-1273; Biological: Continue IS (B cell depletion therapy)
- Cohort C, Arm C2: BNT162b2 + Continue IS (B cell depletion therapy) (Experimental): Adult participants taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will receive an additional dose of the Pfizer-BioNTech COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: BNT162b2; Biological: Continue IS (B cell depletion therapy)
- Cohort C, Arm C3: Ad26.COV2.S + Continue IS (B cell depletion therapy) (Experimental): Arm closed, effective protocol version 3.0. Adult participants taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will receive the Janssen COVID-19 vaccine booster (1 dose) and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Ad26.COV2.S; Biological: Continue IS (B cell depletion therapy)
- Cohort D, Arm D1: Ad26.COV2.S + Withhold IS (MMF or MPA) (Experimental): Arm closed, effective protocol version 4.0. Adult participants who previously received an mRNA vaccine and who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Janssen COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Ad26.COV2.S; Drug: Withhold IS (MMF or MPA)
- Cohort D, Arm D2: Alternative mRNA Vaccine + Withhold IS (MMF or MPA) (Experimental): Adult participants who previously received an mRNA vaccine and who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of an alternative COVID-19 vaccine, per protocol instruction. Beginning with version 6.0 of the protocol, bivalent versions of the mRNA vaccines, Moderna and Pfizer-BioNTech COVID-19 vaccines, replaced original monovalent versions.
  Interventions: Biological: BNT162b2; Drug: Withhold IS (MMF or MPA); Biological: Moderna mRNA-1273, Bivalent; Biological: BNT162b2, Bivalent
- Cohort D, Arm D3: Moderna mRNA-1273 + Withhold IS (MMF or MPA) (Experimental): Adult participants who previously received the Janssen COVID-19 vaccine and who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Moderna COVID-19 vaccine, per protocol instruction. Beginning with version 6.0 of the protocol, bivalent versions of the mRNA vaccines, Moderna and Pfizer-BioNTech COVID-19 vaccines, replaced original monovalent versions.
  Interventions: Drug: Withhold IS (MMF or MPA); Biological: Moderna mRNA-1273, Bivalent
- Cohort E, Arm E1: Ad26.COV2.S + Withhold IS (MTX) (Experimental): Arm closed, effective protocol version 4.0. Adult participants who previously received an mRNA vaccine and who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Janssen COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Ad26.COV2.S; Drug: Withhold IS (MTX)
- Cohort E, Arm E2: Alternative mRNA Vaccine + Withhold IS (MTX) (Experimental): Adult participants who previously received an mRNA vaccine and who are taking methotrexate (without additional B cell depleting medications or MMF/MPA) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of an alternative COVID-19 vaccine, per protocol instruction. Beginning with version 6.0 of the protocol, bivalent versions of the mRNA vaccines, Moderna and Pfizer-BioNTech COVID-19 vaccines, replaced original monovalent versions.
  Interventions: Drug: Withhold IS (MTX); Biological: Moderna mRNA-1273, Bivalent; Biological: BNT162b2, Bivalent
- Cohort E, Arm E3: Moderna mRNA-1273 + Withhold IS (MTX) (Experimental): Adult participants who previously received the Janssen COVID-19 vaccine and who are taking methotrexate (without additional B cell depleting medications or MMF/MPA) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Moderna COVID-19 vaccine, per protocol instruction. Beginning with version 6.0 of the protocol, bivalent versions of the mRNA vaccines, Moderna and Pfizer-BioNTech COVID-19 vaccines, replaced original monovalent versions.
  Interventions: Drug: Withhold IS (MTX); Biological: Moderna mRNA-1273, Bivalent
- Cohort F, Arm F1: Ad26.COV2.S + Withhold IS (B cell depletion therapy) (Experimental): Arm closed, effective protocol version 4.0. Adult participants who previously received an mRNA vaccine and who are taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will continue to take their prescribed BCDTs without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX ) before and after receiving a dose of the Janssen COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Ad26.COV2.S; Drug: Withhold IS (B cell depletion therapy)
- Cohort F, Arm F2: Alternative mRNA Vaccine + Withhold IS (B cell depletion therapy) (Experimental): Adult participants who previously received an mRNA vaccine and who are taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will continue to take their prescribed BCDTs without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the alternative COVID-19 vaccine, per protocol instruction. Beginning with version 6.0 of the protocol, bivalent versions of the mRNA vaccines, Moderna and Pfizer-BioNTech COVID-19 vaccines, replaced original monovalent versions.
  Interventions: Drug: Withhold IS (B cell depletion therapy); Biological: Moderna mRNA-1273, Bivalent; Biological: BNT162b2, Bivalent
- Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (B cell depletion therapy) (Experimental): Adult participants who previously received the Janssen COVID-19 vaccine and who are taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will continue to take their prescribed BCDTs without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Moderna COVID-19 vaccine, per protocol instruction. Beginning with version 6.0 of the protocol, bivalent versions of the mRNA vaccines, Moderna and Pfizer-BioNTech COVID-19 vaccines, replaced original monovalent versions.
  Interventions: Drug: Withhold IS (B cell depletion therapy); Biological: Moderna mRNA-1273, Bivalent
- Cohort D, Arm D4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (MMF or MPA) (Experimental): Adult participants who previously received an mRNA vaccine and who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Sanofi-GSK COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Monovalent [B.1.351] CoV2 preS dTM-AS03; Drug: Withhold IS (MMF or MPA)
- Cohort E, Arm E4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (MTX) (Experimental): Adult participants who previously received an mRNA vaccine and who are taking methotrexate (without additional B cell depleting medications or MMF/MPA) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Sanofi-GSK COVID-19 vaccine, per protocol instruction.
  Interventions: Biological: Monovalent [B.1.351] CoV2 preS dTM-AS03; Drug: Withhold IS (MTX)
- Cohort F, Arm F4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (B cell depletion therapy) (Experimental): Adult participants who previously received an mRNA vaccine and who are taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will continue to take their prescribed BCDTs without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Sanofi-GSK COVID-19 vaccine, per protocol instruction
  Interventions: Biological: Monovalent [B.1.351] CoV2 preS dTM-AS03; Drug: Withhold IS (B cell depletion therapy)
- Cohort A, Arm A1P: Moderna mRNA-1273, Bivalent + Continue IS (MMF or MPA) (Experimental): Pediatric participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will receive an additional dose of the Moderna COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Drug: Continue IS (MMF or MPA); Biological: Moderna mRNA-1273, Bivalent
- Cohort A, Arm A2P: BNT162b2, Bivalent + Continue IS (MMF or MPA) (Experimental): Pediatric participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will receive an additional dose of the Pfizer-BioNTech COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Drug: Continue IS (MMF or MPA); Biological: BNT162b2, Bivalent
- Cohort A, Arm A4P: Moderna mRNA-1273, Bivalent + Withhold IS (MMF or MPA) (Experimental): Pediatric participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MMF or MPA); Biological: Moderna mRNA-1273, Bivalent
- Cohort A, Arm A5P: BNT162b2, Bivalent + Withhold IS (MMF or MPA) (Experimental): Pediatric participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Pfizer-BioNTech COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MMF or MPA); Biological: BNT162b2, Bivalent
- Cohort B, Arm B1P: Moderna mRNA-1273, Bivalent + Continue IS (MTX) (Experimental): Pediatric participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will receive an additional dose of the Moderna COVID-19 vaccine booster and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Drug: Continue IS (MTX); Biological: Moderna mRNA-1273, Bivalent
- Cohort B, Arm B2P: BNT162b2, Bivalent + Continue IS (MTX) (Experimental): Pediatric participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will receive an additional dose of the Pfizer-BioNTech COVID-19 vaccine booster and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Drug: Continue IS (MTX); Biological: BNT162b2, Bivalent
- Cohort B, Arm B4P: Moderna mRNA-1273, Bivalent + Withhold IS (MTX) (Experimental): Pediatric participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MTX); Biological: Moderna mRNA-1273, Bivalent
- Cohort B, Arm B5P: BNT162b2, Bivalent + Withhold IS (MTX) (Experimental): Pediatric participants who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease will withhold their immunosuppressive medications (IS) before and after receiving an additional dose of the Pfizer-BioNTech COVID-19 vaccine booster, per protocol instruction.
  Interventions: Drug: Withhold IS (MTX); Biological: BNT162b2, Bivalent
- Cohort C, Arm C1P: Moderna mRNA-1273, Bivalent + Continue IS (B cell depletion therapy) (Experimental): Pediatric participants taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will receive an additional dose of the Moderna COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Continue IS (B cell depletion therapy); Biological: Moderna mRNA-1273, Bivalent
- Cohort C, Arm C2P: BNT162b2, Bivalent + Continue IS (B cell depletion therapy) (Experimental): Pediatric participants taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will receive an additional dose of the Pfizer-BioNTech COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
  Interventions: Biological: Continue IS (B cell depletion therapy); Biological: BNT162b2, Bivalent
- Cohort D, Arm D1P: BNT162b2, Bivalent + Withhold IS (MMF or MPA) (Experimental): Pediatric participants who previously received the Moderna COVID-19 vaccine and who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Pfizer-BioNTech COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MMF or MPA); Biological: BNT162b2, Bivalent
- Cohort D, Arm D2P: Moderna mRNA-1273, Bivalent + Withhold IS (MMF or MPA) (Experimental): Pediatric participants who previously received the Pfizer-BioNTech COVID-19 vaccine and who are taking MMF or MPA (without additional B cell depleting medications or MTX) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MMF or MPA); Biological: Moderna mRNA-1273, Bivalent
- Cohort E, Arm E1P: BNT162b2, Bivalent + Withhold IS (MTX) (Experimental): Pediatric participants who previously received the Moderna COVID-19 vaccine and who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Pfizer-BioNTech COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MTX); Biological: BNT162b2, Bivalent
- Cohort E, Arm E2P: Moderna mRNA-1273, Bivalent + Withhold IS (MTX) (Experimental): Pediatric participants who previously received the Pfizer-BioNTech COVID-19 vaccine and who are taking methotrexate (without additional B cell depleting medications or MMF/ MPA) for management of their underlying autoimmune disease, will withhold their immunosuppressive medications (IS) before and after receiving a dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (MTX); Biological: Moderna mRNA-1273, Bivalent
- Cohort F, Arm F1P: BNT162b2, Bivalent + Withhold IS (B cell depletion therapy) (Experimental): Pediatric participants who previously received the Moderna COVID-19 vaccine and who are taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will continue to take their prescribed BCDTs without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Pfizer-BioNTech COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (B cell depletion therapy); Biological: BNT162b2, Bivalent
- Cohort F, Arm F2P: Moderna mRNA-1273, Bivalent + Withhold IS (B cell depletion therapy) (Experimental): Pediatric participants who previously received the Pfizer-BioNTech COVID-19 vaccine and who are taking B cell depletion medication(s) for management of their underlying autoimmune disease, regardless of whether they are also taking MMF or MTX, will continue to take their prescribed BCDTs without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Moderna COVID-19 vaccine, per protocol instruction.
  Interventions: Drug: Withhold IS (B cell depletion therapy); Biological: Moderna mRNA-1273, Bivalent

INTERVENTIONS:
Biological: Moderna mRNA-1273 — Administration: One dose administered intramuscularly.
  Other Names: mRNA-1273 vaccine (Moderna); Moderna COVID-19 Vaccine; SARS-CoV-2 RNA vaccine; COVID-19 vaccine
  Arms: Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA); Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA); Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX); Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX); Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (B cell depletion therapy)
Biological: BNT162b2 — Administration: One dose administered intramuscularly.
  Other Names: mRNA-1273 vaccine (Pfizer/BioNTech); SARS-CoV-2 RNA vaccine; Pfizer-BioNTech COVID-19 vaccine
  Arms: Cohort A, Arm A2: BNT162b2 + Continue IS (MMF or MPA); Cohort A, Arm A5: BNT162b2 + Withhold IS (MMF or MPA); Cohort B, Arm B2: BNT162b2 + Continue IS (MTX); Cohort B, Arm B5: BNT162b2 + Withhold IS (MTX); Cohort C, Arm C2: BNT162b2 + Continue IS (B cell depletion therapy); Cohort D, Arm D2: Alternative mRNA Vaccine + Withhold IS (MMF or MPA)
Biological: Ad26.COV2.S — Administration: One dose administered intramuscularly.
  Other Names: Janssen COVID-19 Vaccine; JNJ-78436735
  Arms: Cohort A, Arm A3: Ad26.COV2.S + Continue IS (MMF or MPA); Cohort A, Arm A6: Ad26.COV2.S + Withhold IS (MMF or MPA); Cohort B, Arm B3: Ad26.COV2.S + Continue IS (MTX); Cohort B, Arm B6: Ad26.COV2.S + Withhold IS (MTX); Cohort C, Arm C3: Ad26.COV2.S + Continue IS (B cell depletion therapy); Cohort D, Arm D1: Ad26.COV2.S + Withhold IS (MMF or MPA); Cohort E, Arm E1: Ad26.COV2.S + Withhold IS (MTX); Cohort F, Arm F1: Ad26.COV2.S + Withhold IS (B cell depletion therapy)
Drug: Continue IS (MMF or MPA) — Participants continue to take their immunosuppressive (IS) medications for management of their autoimmune disease without alterations in schedule and dosing.
  Other Names: immunosuppressive medication; mycophenolate mofetil; MMF; CellCept®; mycophenolic acid; MPA
  Arms: Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA); Cohort A, Arm A1P: Moderna mRNA-1273, Bivalent + Continue IS (MMF or MPA); Cohort A, Arm A2: BNT162b2 + Continue IS (MMF or MPA); Cohort A, Arm A2P: BNT162b2, Bivalent + Continue IS (MMF or MPA); Cohort A, Arm A3: Ad26.COV2.S + Continue IS (MMF or MPA)
Drug: Continue IS (MTX) — Participants continue to take their immunosuppressive (IS) medications for management of their autoimmune disease without alterations in schedule and dosing.
  Other Names: methotrexate; MTX
  Arms: Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX); Cohort B, Arm B1P: Moderna mRNA-1273, Bivalent + Continue IS (MTX); Cohort B, Arm B2: BNT162b2 + Continue IS (MTX); Cohort B, Arm B2P: BNT162b2, Bivalent + Continue IS (MTX); Cohort B, Arm B3: Ad26.COV2.S + Continue IS (MTX)
Biological: Continue IS (B cell depletion therapy) — Participants will continue to take their prescribed immunosuppressive (IS) medications without alterations in schedule and dosing.
  Other Names: mAbs targeting CD19 or CD20; anti-BAFF mAb
  Arms: Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (B cell depletion therapy); Cohort C, Arm C1P: Moderna mRNA-1273, Bivalent + Continue IS (B cell depletion therapy); Cohort C, Arm C2: BNT162b2 + Continue IS (B cell depletion therapy); Cohort C, Arm C2P: BNT162b2, Bivalent + Continue IS (B cell depletion therapy); Cohort C, Arm C3: Ad26.COV2.S + Continue IS (B cell depletion therapy)
Biological: Monovalent [B.1.351] CoV2 preS dTM-AS03 — One dose administered intramuscularly
  Other Names: Sanofi-GSK COVID-19 Vaccine
  Arms: Cohort D, Arm D4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (MMF or MPA); Cohort E, Arm E4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (MTX); Cohort F, Arm F4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (B cell depletion therapy)
Drug: Withhold IS (MMF or MPA) — Participants withhold their cohort-defining immunosuppressive (IS) medications for management of their autoimmune disease before and after the additional vaccine dose per protocol instructions.
  Other Names: immunosuppressive medication; mycophenolate mofetil; MMF; CellCept®; mycophenolic acid; MPA
  Arms: Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA); Cohort A, Arm A4P: Moderna mRNA-1273, Bivalent + Withhold IS (MMF or MPA); Cohort A, Arm A5: BNT162b2 + Withhold IS (MMF or MPA); Cohort A, Arm A5P: BNT162b2, Bivalent + Withhold IS (MMF or MPA); Cohort A, Arm A6: Ad26.COV2.S + Withhold IS (MMF or MPA); Cohort D, Arm D1: Ad26.COV2.S + Withhold IS (MMF or MPA); Cohort D, Arm D1P: BNT162b2, Bivalent + Withhold IS (MMF or MPA); Cohort D, Arm D2: Alternative mRNA Vaccine + Withhold IS (MMF or MPA); Cohort D, Arm D2P: Moderna mRNA-1273, Bivalent + Withhold IS (MMF or MPA); Cohort D, Arm D3: Moderna mRNA-1273 + Withhold IS (MMF or MPA); Cohort D, Arm D4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (MMF or MPA)
Drug: Withhold IS (MTX) — Participants withhold their cohort-defining immunosuppressive (IS) medications for management of their autoimmune disease before and after the additional vaccine dose per protocol instructions.
  Other Names: methotrexate; MTX
  Arms: Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX); Cohort B, Arm B4P: Moderna mRNA-1273, Bivalent + Withhold IS (MTX); Cohort B, Arm B5: BNT162b2 + Withhold IS (MTX); Cohort B, Arm B5P: BNT162b2, Bivalent + Withhold IS (MTX); Cohort B, Arm B6: Ad26.COV2.S + Withhold IS (MTX); Cohort E, Arm E1: Ad26.COV2.S + Withhold IS (MTX); Cohort E, Arm E1P: BNT162b2, Bivalent + Withhold IS (MTX); Cohort E, Arm E2: Alternative mRNA Vaccine + Withhold IS (MTX); Cohort E, Arm E2P: Moderna mRNA-1273, Bivalent + Withhold IS (MTX); Cohort E, Arm E3: Moderna mRNA-1273 + Withhold IS (MTX); Cohort E, Arm E4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (MTX)
Drug: Withhold IS (B cell depletion therapy) — Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX ) before and after the additional vaccine dose per protocol instructions. Participants will continue to take their prescribed BCDTs without alterations in schedule and dosing.
  Other Names: mAbs targeting CD19 or CD20; anti-BAFF mAb
  Arms: Cohort F, Arm F1: Ad26.COV2.S + Withhold IS (B cell depletion therapy); Cohort F, Arm F1P: BNT162b2, Bivalent + Withhold IS (B cell depletion therapy); Cohort F, Arm F2: Alternative mRNA Vaccine + Withhold IS (B cell depletion therapy); Cohort F, Arm F2P: Moderna mRNA-1273, Bivalent + Withhold IS (B cell depletion therapy); Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (B cell depletion therapy); Cohort F, Arm F4: Monovalent [B.1.351] CoV2 preS dTM-AS03 + Withhold IS (B cell depletion therapy)
Biological: Moderna mRNA-1273, Bivalent — Administration: One dose administered intramuscularly.
  Other Names: mRNA-1273 vaccine (Moderna), Bivalent; Moderna COVID-19 Vaccine, Bivalent; SARS-CoV-2 RNA vaccine, Bivalent; COVID-19 vaccine, Bivalent
  Arms: Cohort A, Arm A1P: Moderna mRNA-1273, Bivalent + Continue IS (MMF or MPA); Cohort A, Arm A4P: Moderna mRNA-1273, Bivalent + Withhold IS (MMF or MPA); Cohort B, Arm B1P: Moderna mRNA-1273, Bivalent + Continue IS (MTX); Cohort B, Arm B4P: Moderna mRNA-1273, Bivalent + Withhold IS (MTX); Cohort C, Arm C1P: Moderna mRNA-1273, Bivalent + Continue IS (B cell depletion therapy); Cohort D, Arm D2: Alternative mRNA Vaccine + Withhold IS (MMF or MPA); Cohort D, Arm D2P: Moderna mRNA-1273, Bivalent + Withhold IS (MMF or MPA); Cohort D, Arm D3: Moderna mRNA-1273 + Withhold IS (MMF or MPA); Cohort E, Arm E2: Alternative mRNA Vaccine + Withhold IS (MTX); Cohort E, Arm E2P: Moderna mRNA-1273, Bivalent + Withhold IS (MTX); Cohort E, Arm E3: Moderna mRNA-1273 + Withhold IS (MTX); Cohort F, Arm F2: Alternative mRNA Vaccine + Withhold IS (B cell depletion therapy); Cohort F, Arm F2P: Moderna mRNA-1273, Bivalent + Withhold IS (B cell depletion therapy); Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (B cell depletion therapy)
Biological: BNT162b2, Bivalent — Administration: One dose administered intramuscularly.
  Other Names: mRNA-1273 vaccine (Pfizer/BioNTech), Bivalent; SARS-CoV-2 RNA vaccine, Bivalent; Pfizer-BioNTech COVID-19 vaccine, Bivalent
  Arms: Cohort A, Arm A2P: BNT162b2, Bivalent + Continue IS (MMF or MPA); Cohort A, Arm A5P: BNT162b2, Bivalent + Withhold IS (MMF or MPA); Cohort B, Arm B2P: BNT162b2, Bivalent + Continue IS (MTX); Cohort B, Arm B5P: BNT162b2, Bivalent + Withhold IS (MTX); Cohort C, Arm C2P: BNT162b2, Bivalent + Continue IS (B cell depletion therapy); Cohort D, Arm D1P: BNT162b2, Bivalent + Withhold IS (MMF or MPA); Cohort D, Arm D2: Alternative mRNA Vaccine + Withhold IS (MMF or MPA); Cohort E, Arm E1P: BNT162b2, Bivalent + Withhold IS (MTX); Cohort E, Arm E2: Alternative mRNA Vaccine + Withhold IS (MTX); Cohort F, Arm F1P: BNT162b2, Bivalent + Withhold IS (B cell depletion therapy); Cohort F, Arm F2: Alternative mRNA Vaccine + Withhold IS (B cell depletion therapy)

SUMMARY:
This is a randomized, multi-site, adaptive, open-label clinical trial comparing the immune response to different additional doses of COVID-19 vaccine in participants with autoimmune disease requiring IS medications. All study participants will have negative serologic or suboptimal responses (defined as a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL) or a low immune response (defined as a Roche Elecsys® Anti-SARS-CoV-2 S result >200 U/ml and ≤2500 U/mL) to their previous doses of COVID-19 vaccine.

The study will focus on 5 autoimmune diseases in adults:

* Systemic Lupus Erythematosus (SLE)
* Rheumatoid Arthritis (RA)
* Multiple Sclerosis (MS)
* Systemic Sclerosis (SSc), and
* Pemphigus.

This study will focus on 4 autoimmune diseases in pediatric participants:

* Systemic Lupus Erythematosus (SLE)
* Juvenile Idiopathic Arthritis (JIA)
* Pediatric-Onset Multiple Sclerosis (POMS)
* Juvenile Dermatomyositis (JDM)

DETAILED DESCRIPTION:
Adult Population:

Stage 1 of this trial will enroll up to a maximum of 900 adult study participants (up to 60 participants per arm).

Participants will be assigned to one of 3 cohorts based on their IS regimens:

* Cohort A: Receipt of MMF or MPA
* Cohort B: Receipt of MTX
* Cohort C: Receipt of any BCDT within the past 18 months.

Treatment Arms: Participants in Cohorts A, B, and C will be assigned to receive an additional dose of the same COVID-19 vaccine as their original vaccine series. The trial initially enrolled participants who were vaccinated with the Pfizer-BioNTech COVID-19 Vaccine, the Moderna COVID-19 Vaccine, and the Janssen COVID-19 Vaccine. Update: Arms to receive an additional homologous vaccine dose after an initial Janssen COVID 19 Vaccine were closed to enrollment after the CDC updated its recommendations to express a clinical preference for individuals to receive an mRNA COVID-19 vaccine over the Janssen COVID-19 vaccine. All Adult Stage 1 treatment arms were closed to enrollment on 15 August 2022.

Participants in Cohorts A and B will be randomized into 2 IS medication treatment plans as follows:

* Participants continue to take their cohort-defining IS medications without alterations in schedule and dosing.
* Participants withhold their cohort-defining IS medications before and after the additional homologous vaccine dose per protocol instructions.

A participant will be enrolled in the study for a maximum of approximately 13 months.

Stage 2 of this trial will include up to a maximum of 960 adult study participants (up to 80per arm) with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤2500 U/mL after previous COVID-19 vaccine administration (at least 3 doses of mRNA vaccine(s) or 2 doses of the Janssen COVID-19 Vaccine). Participants will be eligible to receive a dose of an alternative COVID-19 vaccine.

Participants may have received their previous COVID-19 vaccine prior to enrollment in the study ("newly recruited participant"), or they may have received their previous COVID-19 vaccine as a study participant and then (re-) enter into Stage 2 ("rollover participant"). Participants can also roll over into Stage 2 via two pathways:

* Stage 1 participant rolls over to Stage 2
* Stage 2 participant rolls over to a different Stage 2 treatment arm

Participants will be allocated to 1 of 3 cohorts based on their IS regimens:

* Cohort D: Receipt of MMF or MPA
* Cohort E: Receipt of MTX
* Cohort F: Receipt of any BCDT within the past 18 months.

Treatment Arms: Participants in Cohorts D, E, and F will receive a dose of an alternative COVID-19 vaccine compared to their previous COVID-19 vaccine doses. Originally, participants who previously received 3 total doses of a single mRNA vaccine (Moderna COVID-19 Vaccine OR Pfizer- BioNTech COVID-19 Vaccine) received their choice of either the Janssen vector-based COVID-19 vaccine or the other mRNA COVID-19 vaccine, and participants who previously received 2 doses of the Janssen vector based COVID-19 vaccine received the Moderna COVID-19 Vaccine.

Update: Beginning with v4.0 of the protocol, this trial will not utilize the Janssen vector-based COVID-19 vaccine. Participants who previously received 3 total doses of a single mRNA vaccine will receive their choice of an alternative mRNA COVID-19 vaccine or the Sanofi-GSK protein based COVID-19 vaccine. Participants who previously received 4 or more doses of a single mRNA vaccine or 3 or more doses of a mixture mRNA vaccines (Moderna COVID-19 Vaccine AND Pfizer-BioNTech COVID-19 Vaccine, in any order or combination) will receive the Sanofi-GSK protein-based COVID-19 vaccine.

Participants in Cohorts D and E will withhold their cohort-defining IS medications before and after the alternative vaccine dose per protocol instructions. Participants in Cohort F who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications before and after the alternative vaccine dose per protocol instructions.

Visits to assess endpoints will occur at Baseline (Week 0), Week 4 ± 1 week, Week 12 ± 2 weeks, Week 24 ± 2 weeks, Week 36 ± 2 weeks, and Week 48 ± 2 weeks. A participant who is newly recruited to the study for entry into Stage 2 may be on study for up to a maximum of 13 months. A participant who enters Stage 2 after a serologic negative, suboptimal, or low immune response to their Stage 1 vaccine dose may be on study for up to a maximum of 26 months. Rollover participants will discontinue follow-up as part of Stage 1 upon rollover into Stage 2. A participant who rolls over to a different Stage 2 treatment arm 2 after a serologic negative, suboptimal, or low immune response to another Stage 2 vaccine dose may be on study for up to a maximum of 38 months.

Pediatric Population:

Stage 1 in the pediatric portion of this trial will enroll up to a maximum of 800 participants (2-17 years of age) with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤2500 U/mL after receiving an initial COVID-19 vaccine regimen (up to 80participants per arm). Vaccines will be included in this protocol as they receive EUA or approval by FDA for a given age group. Pediatric participants will have 1 of 4 autoimmune diseases: pediatric SLE, juvenile idiopathic arthritis (JIA), juvenile dermatomyositis (JDM), or pediatriconset multiple sclerosis (POMS). Participants will be assigned to 1 of 3 cohorts based on their IS regimens:

* Cohort A: Receipt of MMF or MPA
* Cohort B: Receipt of MTX
* Cohort C: Receipt of any BCDT within the past 18 months.

Treatment Arms: Participants in Cohorts A, B, and C will be assigned to receive an additional dose of the same vaccine as their original vaccine series. Based on FDA EUA status, pediatric participants were initially eligible to receive the Pfizer-BioNTech COVID-19 Vaccine only.

Participants in Cohorts A and B will be randomized into 2 IS medication treatment plans as follows):

* Participants continue to take their cohort-defining IS medications without alterations in schedule and dosing.
* Participants withhold their cohort-defining IS medications before and after the additional homologous vaccine dose per protocol instructions.

A participant will be enrolled in the study for a maximum of approximately 13 months.

Stage 2 of the pediatric portion of this trial will include up to a maximum of 480 pediatric study participants (up to 80 per arm) with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤2500 U/mL after previous COVID-19 vaccine administration (an age-appropriate EUA-authorized or FDA-approved initial COVID-19 vaccine regimen plus 1 additional dose of the same vaccine). All participants (2-17 years of age) who previously received doses of the Pfizer-BioNTech COVID-19 Vaccine are eligible to receive an age-appropriate dose of the Moderna COVID-19 Vaccine. Participants 12 through 17 years of age who previously received doses of the Moderna COVID-19 vaccine are eligible to receive an age-appropriate dose of the Pfizer-BioNTech COVID-19 Vaccine. Participants will be eligible to receive a dose of an alternative COVID-19 vaccine. Participants may have received their previous COVID-19 vaccine as a study participant and then enter into Stage 2 ("rollover participant"), or they may have received their previous COVID-19 vaccine prior to enrollment in the study ("newly recruited participant").

Participants will be allocated to 1 of 3 cohorts based on their IS regimens:

* Cohort D: Receipt of MMF or MPA (± other rheumatic disease medications, including biologics)

  o Participants who are taking MMF or MPA (without additional B cell depleting medications or MTX) will be placed in this cohort.
* Cohort E: Receipt of MTX (± other rheumatic disease medications, including biologics)

  o Participants who are taking MTX (without additional B cell depleting medications or MMF/ MPA) will be placed in this cohort.
* Cohort F: Receipt of B cell depletion therapy within the past 18 months (± other rheumatic disease medications) o Participants taking B cell depletion medications, regardless of whether they are also taking MMF or MTX, will be placed in this cohort.

Treatment Arms: Participants in Cohorts D, E, and F will receive a dose of an alternative COVID-19 vaccine compared to their previous COVID-19 vaccine doses. Participants who previously received age-appropriate doses of a single mRNA vaccine (Moderna COVID-19 Vaccine OR Pfizer-BioNTech COVID-19 Vaccine, as noted above) will receive the other mRNA COVID-19 vaccine.

Beginning with v7.0 of the protocol all vaccines used are bivalent versions replacing original monovalent versions.

Participants in Cohorts D and E will withhold their cohort-defining IS medications before and after the alternative vaccine dose per protocol instructions (see Section 7.1.1 Protocol-mandated Medications).

Participants in Cohort F who are taking MMF, MPA, or MTX in addition to B cell depletion therapies (BCDTs) will withhold these medications before and after the alternative vaccine dose per protocol instruction.

A participant who enters Stage 2 after a serologic negative, suboptimal, or low immune response to their Stage 1 vaccine dose may be on study for up to a maximum of 26 months. Rollover participants will discontinue follow-up as part of Stage 1 upon rollover into Stage 2. A participant who is newly recruited to the study for entry into Stage 2 may be on study for up to a maximum of 13 months.

Adaptive Design

An adaptive design will be employed such that cohorts and arms defined by additional vaccine doses and IS treatment plans may be added or modified based on emerging data from existing and new FDA Emergency Use Authorization (EUA) or approvals of COVID-19 vaccines:

* New cohorts may be defined based on changes in the medication groups if it becomes obvious that certain medications are highly associated with suboptimal or low immune serologic response to initial COVID-19 vaccine regimen.
* Cohorts may limit or expand the autoimmune diseases that are eligible to be included in the clinical trial and may include expansion cohorts of underrepresented diseases.
* New cohorts may include participants whose antibody response falls to suboptimal or low immune levels over time.
* Based upon timing of the FDA EUA authorization for children of each of the COVID-19 vaccines used in this trial, the age range of the inclusion criteria may be expanded.
* Allocation or randomization to treatment with new COVID-19 vaccines may be incorporated into the design when the products become available.
* Identification of additional strategies to enhance vaccine responsiveness in autoimmune diseases, including a temporary switch of immunomodulatory medications.

ELIGIBILITY:
General Adult Inclusion Criteria:

1. Willing and able to sign informed consent 2. Documented full COVID-19 vaccination (CDC card or documentation in medical records) that was completed at least 4 weeks prior and no more than 52 weeks prior to the Stage 1 Screening visit, or if participating in Stage 2, no more than 48 weeks prior to the Stage 2 Screening visit.

General Exclusion Criteria 2. History of severe allergic reaction to the initial COVID-19 vaccine regimen, to any component of any of the COVID-19 vaccines, or to polyethylene glycol (PEG).

3. New diagnosis of malignancy that will require chemotherapy or immunotherapy, or ongoing treatment for a malignancy with chemotherapy or immunotherapy.

4. Active disease (per the Investigator's decision) resulting in inability to hold the IS therapy in the MMF/MPA or MTX arms of the study.

a. The potential impact of temporarily holding medication for participants with a recent mild disease flare within 4 weeks should be carefully considered.

5. Active disease during the Screening period resulting in:

1. An increase/addition of any IS medications, or
2. A suggestion of MS relapse per the investigator. 6. Recent or current SARS-CoV-2 infection defined as:

<!-- -->

1. Documented SARS-CoV-2 infection in the past 30 days (from the day the participant is diagnosed by positive test to Screening).
2. Positive result on a molecular COVID-19 test at Screening. 8. Inflammatory myocarditis/pericarditis within 6 weeks of any COVID-19 vaccine doses.

   9. Participants with active, ongoing chronic infections. Note: Participants are permitted to be on chronic prophylactic antimicrobial therapy. Adults with evidence of HIV, Hepatitis B indicated by surface antigen, and Hepatitis C indicated by anti-hepatitis C antibody positivity will be excluded. If an adult is negative for Hepatitis C viral load at Screening, he/she will be eligible to participate.

   10. Participants with common variable immunodeficiency disease, as well as any participants currently receiving immune globulin replacement therapy. Note: Pediatric participants on IVIG therapeutically may enter the study provided they have sufficiently quiet disease that they can withhold their IVIG from 8 weeks prior to the Screening visit through 4 weeks after vaccination.

   11. Participants who received licensed or investigational monoclonal antibodies or plasma products directed against SARS-CoV-2 within 30 days of Screening.

   12. Participants who have received any live vaccines within 2 months of the anticipated study vaccine dose or who will have need of a live vaccine at any time during the study.

   13. Currently pregnant or breastfeeding (For pediatric participants postmenarchal females must have a negative urine pregnancy test at Screening).

   15. Hemoglobin (Hgb) <8.0 g/dL (80 g/L) 16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

   17. Other investigational chemical agent within 30 days or other investigational biologic agent within 8 weeks or 5 half-lives (whichever is longer) of Screening.

   18. Concurrent treatment with cyclophosphamide. Adult participants taking cladribine, alemtuzumab, or mitoxantrone will also be excluded.

   19. Participants currently on any type of dialysis, or who have received a solid organ transplant.

   20. Prisoners or participants who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

   21. Taking both MMF/MPA and MTX. 22. Receiving other investigational BCDT as part of a clinical trial within 18 months of Screening, unless drug assignment is known and the participant received an anti-CD20 or CD19 drug.

   23. Participants with active systemic infections who have received systemic antimicrobials within the 14 days prior to Screening.

   Adult General Criteria

   Inclusion Criteria:
   1. Individuals 18 years of age or older that meet classification criteria for systemic lupus erythematosus (SLE), systemic sclerosis (SSc), rheumatoid arthritis (RA), multiple sclerosis (MS), or pemphigus
   2. Participants must meet the 2019 ACR/EULAR or 2012 SLICC classification criteria for SLE, the 2010 ACR/EULAR classification criteria for RA, the 2013 EULAR/ACR classification criteria for SSc, the 2017 McDonald criteria for MS, and the international consensus criteria for pemphigus.

<!-- -->

1. If a participant has been diagnosed with more than one autoimmune disease, the participant will be assessed based on the disease that is selected for study entry 6. Must be currently taking one of the following IS medications with or without additional disease-related medications: MMF (minimum of 1000 mg per day)/MPA (minimum of 720 mg per day), MTX (minimum of 7.5mg per week), or B cell depleting agents within the past 18 months (such as rituximab, ocrelizumab, ofatumumab).

<!-- -->

1. If taking MMF/MPA or MTX, the participant must have initiated therapy at least 8 weeks prior to randomization and be taking the same medications (regardless of dose) as at the time of the initial COVID-19 vaccine regimen. Note: Participants who withheld their IS medications around their initial vaccinations are eligible to participate.
2. If enrolling in the BCDT cohort, the participant must have received an anti-CD20 or an anti-CD19 BCDT in the past 18 months.

   7. No changes in background IS medications, including MMF/MPA or MTX, in the 4 weeks prior to Screening, excluding the following:

<!-- -->

1. HCQ,
2. Intraarticular steroids,
3. The addition of prednisone at ≤10mg per day or prednisone at any dose when given for ≤3 days, and
4. Corticosteroid bursts for non-autoimmune disease-related conditions, such as asthma or COPD, are permitted.

   Adult General Exclusion Criterion 1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.

   14. Adult female participants who are planning a pregnancy during the course of the trial.

   Adult Stage 1-Specific Inclusion Criterion 5. Negative or suboptimal serologic response to initial COVID-19 vaccine regimen, defined as an Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL, at Screening visit.

<!-- -->

1. Initial COVID-19 vaccine regimen is defined as either:

i.2 doses of the Pfizer-BioNTech COVID-19 Vaccine ii. 2 doses of the Moderna COVID-19 Vaccine

Adult Stage 1-Specific Exclusion Criterion 7. Receipt of a COVID-19 vaccine booster prior to Screening with the Moderna COVID-19 Vaccine, Pfizer-BioNTech COVID-19 Vaccine, or Janssen COVID-19 Vaccine.

Adult Stage 2 (Newly Recruited)-Specific Inclusion Criteria 2. History of severe allergic reaction to the COVID-19 vaccine, or to any component of the COVID-19 vaccine, that is to be administered in Stage 2, including polysorbate for participants receiving the Sanofi-GSK COVID-19 Vaccine, or to PEG.

5. Negative or suboptimal serologic response to a previous COVID 19 vaccine administration in one of the qualifying regimens, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) negative result or positive result of ≤200 U/mL, or a low immune response, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) result of ≤2500 U/mL, within 4 weeks of the Stage 2 Baseline/Week 0 visit. The regimens of COVID-19 vaccination that qualify are as follows:

1. 3 doses of the Pfizer-BioNTech COVID-19 Vaccine
2. 3 doses of the Moderna COVID-19 Vaccine
3. 2 doses of the Janssen COVID-19 Vaccine
4. 4 or more doses of a single mRNA vaccine (Pfizer-BioNTech COVID-19 Vaccine OR Moderna COVID-19 Vaccine)
5. 3 or more doses of a mixture of mRNA vaccines (Pfizer-BioNTech COVID-19 Vaccine OR Moderna COVID-19 Vaccine)

Adult Stage 2 (Newly Recruited)-Specific Exclusion Criteria:

7. Receipt of a mixture of Janssen COVID-19 vaccines and mRNA COVID-19 vaccines (in any order or combination) prior to Stage 2 Screening.

Adult Stage 2 (Rollover)-Specific Inclusion Criteria:

Individuals who were previously enrolled in Adult Stage 1 or Adult Stage 2 will have met some inclusion and exclusion criteria at that time. Only a subset of the criteria for (re-)entering Adult Stage 2 will be assessed in rollover participants at the time of screening for Stage 2.

Individuals who meet all of the following criteria are eligible to (re )enter Adult Stage 2:

2. History of severe allergic reaction to the COVID-19 vaccine, or to any component of the COVID-19 vaccine, that is to be administered in Stage 2, including polysorbate for participants receiving the Sanofi-GSK COVID-19 Vaccine, or to PEG.

5. Negative or suboptimal serologic response to a previous COVID 19 vaccine administration in one of the qualifying regimens, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) negative result or positive result of ≤200 U/mL, or a low immune response, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) result of ≤2500 U/mL, within 4 weeks of the Stage 2 Baseline/Week 0 visit. The regimens of COVID-19 vaccination that qualify are as follows:

a. 3 doses of the Pfizer-BioNTech COVID-19 Vaccine b. 3 doses of the Moderna COVID-19 Vaccine c. 2 doses of the Janssen COVID-19 Vaccine d. 4 doses of a combination of mRNA vaccines (i.e., Pfizer-BioNTech COVID-19 Vaccine, Moderna COVID-19 Vaccine)

General Pediatric Inclusion Criteria

1. Individuals 2-17 years of age that meet classification criteria for SLE, JIA, POMS, or JDM. Note: Juvenile idiopathic arthritis includes the following conditions: polyarticular JIA (both RF + and -), oligoarticular persistent and oligoarticular extended JIA, psoriatic arthritis, and enthesitis related JIA.

   1. Participants must meet the 2017 EULAR/ACR classification criteria for adult and juvenile idiopathic inflammatory myopathies and their major subgroups, the International League of Associations for Rheumatology (ILAR) classification for JIA, the 2017 McDonald criteria for MS, or the Bohan and Peter criteria or the 2017 EULAR/ACR classification criteria for JDM.
   2. If a participant has been diagnosed with more than one autoimmune disease, the participant will be assessed based on the disease that is selected for study entry.
2. Parents/guardians of all pediatric participants and participants ages 14 - 17 must be willing and able to sign informed consent. Participants ages 7-13 must be willing and able to sign assent.

5. Must be currently taking one of the following IS medications with or without additional disease-related medications: MMF (minimum of 250 mg per day)/MPA (minimum of 360 mg per day), MTX (minimum of 5 mg per week), or B cell depleting agents within the past 18 months (such as rituximab, ocrelizumab, or ofatumumab).

1. If taking MMF/MPA or MTX, the participant must have initiated therapy at least 8 weeks prior to randomization and be taking the same medications (regardless of dose) as at the time of the initial COVID-19 vaccine regimen. Note: Participants who withheld their IS medications around their initial vaccinations are eligible to participate.
2. If enrolling in the BCDT cohort, participant must have received an anti-CD20 or an anti-CD19 BCDT in the past 18 months.

   6. No changes in background IS medications, including MMF/MPA or MTX, in the 8 weeks prior to Screening, excluding the following:

a. HCQ, b. Intraarticular steroids, c. The addition of prednisone at <0.15mg/kg/dose per day or prednisone at any dose when given for ≤3 days, and d. Corticosteroid bursts for non-autoimmune disease-related conditions, such as asthma or COPD, are permitted

General Pediatric Exclusion Criteria 1. Inability or unwillingness of a participant to give assent or of a parent/guardian to give written informed consent, or of either to comply with study protocol.

Pediatric Stage 1-Specific Inclusion Criteria:

4. Negative or suboptimal serologic response to initial EUA-authorized or FDA-approved COVID-19 vaccine doses, defined as an Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL, or a low immune response, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) result of ≤2500 U/mL, within 4 weeks of the Stage 1 Baseline/Week 0 visit

Initial COVID-19 vaccine regimen is defined as:

i. Pfizer-BioNTech COVID-19 Vaccine (2 through 4 years of age): 3 age-appropriate doses ii. Pfizer-BioNTech COVID-19 Vaccine (5 through 17 years of age): 2 age-appropriate doses iii. Moderna COVID-19 Vaccine (2 through 17 years of age): 2 age-appropriate doses.

Pediatric Stage 1-Specific Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for randomization/allocation as participants in the pediatric portion of the study:

7. Receipt of a COVID-19 vaccine booster prior to Screening.

Pediatric Stage 2 (Newly Recruited)-Specific Inclusion Criteria 5. Negative or suboptimal serologic response to homologous doses of COVID-19 vaccine in one of the qualifying regimens, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) negative result or positive result of ≤200 U/mL, or a low immune response, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) result of ≤2500 U/mL, within 4 weeks of the Stage 2 Baseline/Week 0 visit. The regimens of COVID-19 vaccination that qualify are as follows: a. Pfizer-BioNTech COVID-19 Vaccine (2 through 5 years of age): 4 full, age-appropriate doses of the Pfizer-BioNTech COVID-19 Vaccine b. Pfizer-BioNTech COVID-19 Vaccine (5 through 17 years old): 3 full, age-appropriate doses of the Pfizer-BioNTech COVID-19 Vaccine Note: Participants who are 5 years old and previously received the Pfizer-BioNTech COVID-19 Vaccine may have received either age-appropriate regimen.

c. Moderna COVID-19 Vaccine (12 through 17 years of age): 3 full, age-appropriate doses of the Moderna COVID-19 Vaccine

Pediatric Stage 2 (Newly Recruited)-Specific Exclusion Criteria:

7. Receipt of an additional heterologous COVID-19 vaccine dose prior to Stage 2 Screening, i.e., a participant cannot have received a mixture of mRNA vaccines.

Pediatric Stage 2 (Rollover)-Specific Inclusion Criteria:

5. Negative or suboptimal serologic response to a previous COVID-19 vaccine administration in one of the qualifying regimens, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) negative result or positive result of ≤200 U/mL, or a low immune response, defined as an Elecsys® Anti-SARS-CoV-2 S (RBD) result of ≤2500 U/mL, within 4 weeks of the Stage 2 Baseline/Week 0 visit. The regimens of COVID-19 vaccination that qualify are as follows:

1. Pfizer-BioNTech COVID-19 Vaccine (2 through 5 years of age): 4 full, age-appropriate doses of the Pfizer-BioNTech COVID-19 Vaccine
2. Pfizer-BioNTech COVID-19 Vaccine (5 through 17 years old): 3 full, age-appropriate doses of the Pfizer-BioNTech COVID-19 Vaccine Note: Participants who are 5 years old and previously received the Pfizer-BioNTech COVID-19 Vaccine may have received either age-appropriate regimen.
3. Moderna COVID-19 Vaccine (12 through 17 years of age): 3 full, age-appropriate doses of the Moderna COVID-19 Vaccine

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. James, MD, PhD, Study Chair — Arthritis and Clinical Immunology Program, Oklahoma Medical Research Foundation; Meggan C. Mackay, MD, MS, Study Chair — Center of Autoimmune Musculoskeletal and Hematopoietic Diseases, Feinstein Institute for Medical Research; Dinesh Khanna, MBBS, MSc, Study Chair — University of Michigan Health, Michigan Medicine; Amit Bar-Or, MD, FRCP, Study Chair — Center for Neuroinflammation and Neurotherapeutics, Perelman School of Medicine, University of Pennsylvania; Virginia Pascual, MD, Study Chair — Drukier Institute for Children's Health, Weill Cornell Medical College; Stacy Ardoin, MD, Study Chair — Nationwide Children's Hospital Rheumatology Department; Natasha Mckerran Ruth, MD, Study Chair — Medical University of South Carolina, Pediatric Rheumatology; Tracey Wright, MD, Study Chair — UT Southwestern Medical Center, Pediatric Rheumatology
Locations (29):
- United States (29):
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - Yale University School of Medicine: Rheumatology, Allergy & Immunology, New Haven, Connecticut
  - The Emory Clinic: Division of Rheumatology, Atlanta, Georgia
  - Indiana University Medical Center, Riley Hospital for Children, Indianapolis, Indiana
  - Massachusetts General Hospital: Rheumatology, Allergy and Immunology, Center for Immunology and Inflammatory Diseases, Boston, Massachusetts
  - Boston Children's Hospital: Department of Pediatrics, Rheumatology Program, Boston, Massachusetts
  - Brigham & Women's Hospital: Department of Medicine, Rheumatology, Immunology, Boston, Massachusetts
  - University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis: Division of Rheumatology, St Louis, Missouri
  - Feinstein Institute for Medical Research: Center for Autoimmune and Musculoskeletal Diseases, Manhasset, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - New York University Langone Medical Center: Department of Medicine, Division of Rheumatology, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Irving Medical Center: Department of Neurology, Multiple Sclerosis Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - University of North Carolina Children's Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center: Division of Rheumatology and Immunology, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hopspital, Columbus, Ohio
  - Oklahoma Children's Hospital-Pediatrics Specialties Clinic, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation: Arthritis and Clinical Immunology Research Program, Oklahoma City, Oklahoma
  - Temple Health: Rheumatology, Philadelphia, Pennsylvania
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Nexus Research Center, Charleston, South Carolina
  - Medical University of South Carolina, Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - UT Southwestern (Peds), Dallas, Texas
  - University of Texas Houston Medical School: Division of Rheumatology and Clinical Immunogenetics, Houston, Texas
  - Benaroya Research Institute at Virginia Mason: Internal Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Derived] Mackay M, Wagner CA, Pinckney A, Cohen JA, Wallace ZS, Khosroshahi A, Sparks JA, Lord S, Saxena A, Caricchio R, Kim AH, Kamen DL, Koumpouras F, Askanase AD, Smith K, Guthridge JM, Pardo G, Mao-Draayer Y, Macwana S, McCarthy S, Sherman MA, Daneshfar Hamrah S, Veri M, Walker S, York K, Tedeschi SK, Wang J, Dziubla GE, Castro M, Carroll R, Narpala SR, Lin BC, Serebryannyy L, McDermott AB, Barry WT, Goldmuntz E, McNamara J, Payne AS, Bar-Or A, Khanna D, James JA. Prospective SARS-CoV-2 additional vaccination in immunosuppressant-treated individuals with autoimmune diseases in a randomized controlled trial. JCI Insight. 2025 Nov 25:e191266. doi: 10.1172/jci.insight.191266. Online ahead of print. PMID 41289027
- See also: Autoimmunity Centers of Excellence (ACE) — https://www.autoimmunitycenters.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 adult sites and 12 pediatric sites were activated in the United States. 374 adult participants and 9 pediatric participants were screened from August 2021 until April 2023 in Stage 1 and 2 of the trial. Adult arms A3, B3, B6, D1, D3, E1, and E3; Pediatric Stage 1; Pediatric Stage 2 arms D1P, E1P, F1P, and F2P did not randomized/allocate or vaccinate participants. One participant was allocated to Adult arm F1 but was not vaccinated.
Pre-assignment Details: In Stage 2, participants could be newly recruited, consent to rollover from Stage 1 of the trial (43 participants), or could consent to receive a second vaccine (Sanofi-GSK) after receipt of a mRNA vaccine in Stage 2 (19 participants).
Groups:
- Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA): Stage 1 adult participants who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease will receive an additional dose of the Moderna mRNA-1273 COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA): Stage 1 adult participants who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving an additional dose of the Moderna mRNA-1273 COVID-19 vaccine, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA): Stage 1 adult participants who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease will receive an additional dose of the Pfizer-BioNTech (BNT162b2) COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA): Stage 1 adult participants who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving an additional dose of the Pfizer-BioNTech (BNT162b2) COVID-19 vaccine, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA): Stage 1 adult participants who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving an additional dose of the Ad26.COV2.S (Janssen) COVID-19 vaccine, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX): Stage 1 adult participants who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will receive an additional dose of the Moderna mRNA-1273 COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX): Stage 1 adult participants who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving an additional dose of the Moderna mRNA-1273 COVID-19 vaccine (but not for more than 21 days total), per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX): Stage 1 adult participants who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will receive an additional dose of the Pfizer-BioNTech (BNT162b2) COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX): Stage 1 adult participants who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving an additional dose of the Pfizer-BioNTech (BNT162b2) COVID-19 vaccine (but not for more than 21 days total), per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT): Stage 1 adult participants taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate, mycophenolate mofetil or mycophenolic acid, will receive an additional dose of the Moderna mRNA-1273 COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT): Stage 1 adult participants taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate, mycophenolate mofetil or mycophenolic acid, will receive an additional dose of the Pfizer-BioNTech (BNT162b2) COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort C, Arm C3: Janssen + Continue IS (BCDT): Stage 1 adult participants taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate, mycophenolate mofetil or mycophenolic acid, will receive an additional dose of the Ad26.COV2.S (Janssen) COVID-19 vaccine and continue to take their immunosuppressive medications (IS) without alterations in schedule and dosing.
- Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA): Stage 2 adult participants who previously received an mRNA vaccine and who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease, will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving a dose of an alternative COVID-19 vaccine (Moderna mRNA-1273 or Pfizer-BioNTech (BNT162b2)), per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA): Stage 2 adult participants who previously received an mRNA vaccine and who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease, will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving a dose of the Sanofi-GSK (Monovalent [B.1.351] CoV2 preS dTM-AS03) COVID-19 vaccine, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX): Stage 2 adult participants who previously received an mRNA vaccine and who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving a dose of an alternative COVID-19 vaccine (Moderna mRNA-1273 or Pfizer-BioNTech (BNT162b2)), but not for more than 21 days total, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX): Stage 2 adult participants who previously received an mRNA vaccine and who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving a dose of the Sanofi-GSK (Monovalent [B.1.351] CoV2 preS dTM-AS03) vaccine, but not for more than 21 days total, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT): Stage 2 adult participants who previously received an mRNA COVID-19 vaccine and who are taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate (MTX), mycophenolate mofetil (MMF) or mycophenolic acid (MPA), will continue to take their prescribed, cohort-defining, immunosuppressive medications (IS) without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the alternative COVID-19 vaccine (Moderna mRNA-1273 or Pfizer-BioNTech (BNT162b2)), per protocol instruction. MMF and MPA: hold 3 days before and 10 days after vaccine. MTX: hold for at least 7 days before and at least 7 days after vaccine, but not for more than 21 days total.
- Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT): Stage 2 adult participants who previously received the Janssen COVID-19 vaccine and who are taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate (MTX), mycophenolate mofetil (MMF) or mycophenolic acid (MPA), will continue to take their prescribed, cohort-defining, immunosuppressive medications (IS) without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Moderna mRNA-1273 vaccine, per protocol instruction. MMF and MPA: hold 3 days before and 10 days after vaccine. MTX: hold for at least 7 days before and at least 7 days after vaccine, but not for more than 21 days total.
- Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT): Stage 2 adult participants who previously received an mRNA COVID-19 vaccine and who are taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate (MTX), mycophenolate mofetil (MMF) or mycophenolic acid (MPA), will continue to take their prescribed, cohort-defining, immunosuppressive medications (IS) without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Sanofi-GSK (Monovalent [B.1.351] CoV2 preS dTM-AS03) vaccine, per protocol instruction. MMF and MPA: hold 3 days before and 10 days after vaccine. MTX: hold for at least 7 days before and at least 7 days after vaccine, but not for more than 21 days total.
- Cohort F, Arm F1: Janssen + Withhold IS (BCDT): Stage 2 adult participants who previously received an mRNA COVID-19 vaccine and who are taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate (MTX), mycophenolate mofetil (MMF) or mycophenolic acid (MPA), will continue to take their prescribed, cohort-defining, immunosuppressive medications (IS) without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the Ad26.COV2.S (Janssen) vaccine, per protocol instruction. MMF and MPA: hold 3 days before and 10 days after vaccine. MTX: hold for at least 7 days before and at least 7 days after vaccine, but not for more than 21 days total.
- Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA): Stage 2 pediatric participants who previously received the Pfizer-BioNTech COVID-19 vaccine and who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease, will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving a dose of the Moderna mRNA-1273 Bivalent COVID-19 vaccine, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX): Stage 2 pediatric participants who previously received the Pfizer-BioNTech COVID-19 vaccine and who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving a dose of the Moderna mRNA-1273 Bivalent vaccine, but not for more than 21 days total, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
Period: Stage 1
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) | Cohort F, Arm F1: Janssen + Withhold IS (BCDT) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Started | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 5 | 6 | 1 | 2 | 2 | 5 | 9 | 22 | 13 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 4 | 4 | 1 | 1 | 1 | 6 | 2 | 19 | 32 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive vaccine at Week 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Received a SARS-CoV-2 vaccine off study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Rolled over to Stage 2 of the study | 1 | 0 | 3 | 3 | 0 | 1 | 0 | 2 | 0 | 13 | 18 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) | Cohort F, Arm F1: Janssen + Withhold IS (BCDT) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 5 | 0 | 33 | 2 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 24 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive vaccine at Week 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0
Not completed — Received a SARS-CoV-2 vaccine off study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Other reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 Sanofi
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) | Cohort F, Arm F1: Janssen + Withhold IS (BCDT) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 17 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Received a SARS-CoV-2 vaccine off study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized or allocated to study arms for Stage 1, Stage 2 and Stage 2 Sanofi.
Groups:
- Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX): Stage 2 pediatric participants who previously received the Pfizer-BioNTech COVID-19vaccine and who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving a dose of the Moderna mRNA-1273 Bivalent vaccine, but not for more than 21 days total, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Total: Total of all reporting groups
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) | Cohort F, Arm F1: Janssen + Withhold IS (BCDT) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX) | Total
Number analyzed (Participants) | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 9 | 5 | 8 | 6 | 57 | 2 | 20 | 1 | 1 | 1 | 258
Age, Categorical [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 1, Stage 2, and Stage 2 Sanofi.
  Participants
    Stage 1: number analyzed (Participants) | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148
    Stage 1: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 |  |  |  |  |  |  |  |  |  |  | 1
    Stage 1: Between 18 and 65 years | 2 | 2 | 6 | 9 | 2 | 0 | 1 | 6 | 4 | 33 | 40 | 8 |  |  |  |  |  |  |  |  |  |  | 113
    Stage 1: >=65 years | 0 | 0 | 3 | 1 | 0 | 3 | 2 | 5 | 7 | 8 | 4 | 1 |  |  |  |  |  |  |  |  |  |  | 34
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1 | 79
    Stage 2: <=18 years |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  | 1 | 0 |  | 0 | 1 | 1 | 3
    Stage 2: Between 18 and 65 years |  |  |  |  |  |  |  |  |  |  |  |  | 6 |  | 6 |  | 47 | 2 |  | 1 | 0 | 0 | 62
    Stage 2: >=65 years |  |  |  |  |  |  |  |  |  |  |  |  | 3 |  | 2 |  | 9 | 0 |  | 0 | 0 | 0 | 14
    Stage 2 Sanofi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0 | 31
    Stage 2 Sanofi: <=18 years |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
    Stage 2 Sanofi: Between 18 and 65 years |  |  |  |  |  |  |  |  |  |  |  |  |  | 3 |  | 4 |  |  | 16 |  |  |  | 23
    Stage 2 Sanofi: >=65 years |  |  |  |  |  |  |  |  |  |  |  |  |  | 2 |  | 2 |  |  | 4 |  |  |  | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are being reported separately for stage 1, stage 2 and stage 2 Sanofi.
  years
    Stage 1: number analyzed (Participants) | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148
    Stage 1 | 62.0 (2.89) | 41.0 (9.90) | 50.4 (16.34) | 44.7 (13.12) | 59.5 (0.71) | 70.7 (5.69) | 64.7 (17.39) | 62.3 (7.98) | 66.0 (9.96) | 51.3 (14.81) | 45.4 (13.02) | 55.1 (7.15) |  |  |  |  |  |  |  |  |  |  | 51.9 (14.46)
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1 | 79
    Stage 2 |  |  |  |  |  |  |  |  |  |  |  |  | 51.4 (16.46) |  | 62.4 (4.66) |  | 51.1 (13.41) | 54.0 (5.66) |  | 54.0 (NA) — Sample size didn't support displaying the descriptive statistic | 17.0 (NA) — Sample size didn't support displaying the descriptive statistic | 12.0 (NA) — Sample size didn't support displaying the descriptive statistic | 51.5 (14.39)
    Stage 2 Sanofi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0 | 31
    Stage 2 Sanofi |  |  |  |  |  |  |  |  |  |  |  |  |  | 51.6 (19.86) |  | 63.0 (9.19) |  |  | 52.9 (11.09) |  |  |  | 54.7 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 1, Stage 2, and Stage 2 Sanofi.
  Participants
    Stage 1: number analyzed (Participants) | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148
    Stage 1: Female | 2 | 2 | 8 | 9 | 2 | 2 | 3 | 11 | 10 | 27 | 35 | 5 |  |  |  |  |  |  |  |  |  |  | 116
    Stage 1: Male | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 14 | 10 | 4 |  |  |  |  |  |  |  |  |  |  | 32
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1 | 79
    Stage 2: Female |  |  |  |  |  |  |  |  |  |  |  |  | 9 |  | 6 |  | 43 | 1 |  | 1 | 1 | 1 | 62
    Stage 2: Male |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 2 |  | 14 | 1 |  | 0 | 0 | 0 | 17
    Stage 2 Sanofi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0 | 31
    Stage 2 Sanofi: Female |  |  |  |  |  |  |  |  |  |  |  |  |  | 5 |  | 4 |  |  | 19 |  |  |  | 28
    Stage 2 Sanofi: Male |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 2 |  |  | 1 |  |  |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 1, Stage 2, and Stage 2 Sanofi.
  Participants
    Stage 1: number analyzed (Participants) | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148
    Stage 1: Hispanic or Latino | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 5 | 1 |  |  |  |  |  |  |  |  |  |  | 16
    Stage 1: Not Hispanic or Latino | 1 | 2 | 7 | 8 | 1 | 3 | 2 | 11 | 9 | 40 | 40 | 8 |  |  |  |  |  |  |  |  |  |  | 132
    Stage 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1 | 79
    Stage 2: Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  | 0 |  | 4 | 0 |  | 0 | 0 | 0 | 5
    Stage 2: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  | 8 |  | 8 |  | 53 | 2 |  | 1 | 1 | 1 | 74
    Stage 2: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  | 0 | 0 |  | 0 | 0 | 0 | 0
    Stage 2 Sanofi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0 | 31
    Stage 2 Sanofi: Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
    Stage 2 Sanofi: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  |  | 5 |  | 6 |  |  | 20 |  |  |  | 31
    Stage 2 Sanofi: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 1, Stage 2, and Stage 2 Sanofi.
  Participants
    Stage 1: number analyzed (Participants) | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148
    Stage 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 1
    Stage 1: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 |  |  |  |  |  |  |  |  |  |  | 3
    Stage 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Stage 1: Black or African American | 0 | 2 | 3 | 6 | 1 | 0 | 1 | 2 | 3 | 2 | 8 | 2 |  |  |  |  |  |  |  |  |  |  | 30
    Stage 1: White | 2 | 0 | 6 | 3 | 1 | 3 | 1 | 7 | 6 | 38 | 35 | 7 |  |  |  |  |  |  |  |  |  |  | 109
    Stage 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 2
    Stage 1: Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 |  |  |  |  |  |  |  |  |  |  | 3
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1 | 79
    Stage 2: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  | 0 | 0 |  | 0 | 0 | 0 | 0
    Stage 2: Asian |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  | 1 | 0 |  | 0 | 1 | 0 | 2
    Stage 2: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  | 0 | 0 |  | 0 | 0 | 0 | 0
    Stage 2: Black or African American |  |  |  |  |  |  |  |  |  |  |  |  | 2 |  | 0 |  | 6 | 0 |  | 1 | 0 | 0 | 9
    Stage 2: White |  |  |  |  |  |  |  |  |  |  |  |  | 6 |  | 8 |  | 48 | 2 |  | 0 | 0 | 1 | 65
    Stage 2: More than one race |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  | 0 | 0 |  | 0 | 0 | 0 | 0
    Stage 2: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  | 0 |  | 2 | 0 |  | 0 | 0 | 0 | 3
    Stage 2 Sanofi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0 | 31
    Stage 2 Sanofi: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
    Stage 2 Sanofi: Asian |  |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  | 0 |  |  | 1 |  |  |  | 2
    Stage 2 Sanofi: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
    Stage 2 Sanofi: Black or African American |  |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  | 0 |  |  | 2 |  |  |  | 3
    Stage 2 Sanofi: White |  |  |  |  |  |  |  |  |  |  |  |  |  | 3 |  | 6 |  |  | 17 |  |  |  | 26
    Stage 2 Sanofi: More than one race |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
    Stage 2 Sanofi: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |  | 0 |  |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants] — Data are reported separately for Stage 1, Stage 2, and Stage 2 Sanofi.
  Participants
    United States: Stage 1 | 2 | 2 | 9 | 10 | 2 | 3 | 3 | 11 | 11 | 41 | 45 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148
    United States: Stage 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0 | 57 | 2 | 0 | 1 | 1 | 1 | 79
    United States: Stage 2 Sanofi | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6 | 0 | 0 | 20 | 0 | 0 | 0 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percent of Stage 1 Adult Participants Who Have a Protective Antibody Response at Week 4
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center (NIAID-VRC) Meso Scale Discovery (MSD) 3 plex assay (Wu-1 full-length spike, receptor binding domain (RBD), and N proteins). A threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Percentage of participants
  Week 4, Wu-1 Full-Length Spike | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.
  Week 4, Receptor Binding Domain (RBD) | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.

2. Primary Outcome: Percent of Stage 2 Adult Participants Who Have a Protective Antibody Response at Week 4
Description: as for outcome 1
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Percentage of participants
  Week 4, Wu-1 Full-Length Spike | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.
  Week 4, Receptor Binding Domain (RBD) | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.

3. Primary Outcome: Percent of Stage 2 Pediatric Participants Who Have a Protective Antibody Response at Week 4
Description: as for outcome 1
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Percentage of participants
  Week 4, Wu-1 Full-Length Spike | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.
  Week 4, Receptor Binding Domain (RBD) | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial. | NA — Threshold for achieving a protective antibody response was not established for the NIAID VRC MSD assay. The intent was to use a pre-established threshold to define a protective antibody response. However, correlates from previous studies could not be extrapolated to the CoV-2 variants circulating over the entire course of this trial.

4. Secondary Outcome: Percentage of Stage 1 Adult Participants Who Seroconverted
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center Meso Scale Discovery 3 plex assay. For concentrations below the lower limit of detection (LLOD), numeric values equivalent to LLOD/2 were assigned; concentrations above the upper limit of quantification were reported without adjustments. Antibody results collected after a documented COVID-19 infection, monoclonal antibody use, or COVID-19 vaccine given off-study were excluded from the analyses. Participants missing antibody data were considered missing-completely-at-random. Seroconversion was assessed in the subgroup of participants who were anti-COVID-19 antibody negative at Week 0; defined as a result less than or equal to the positive threshold value (spike=10.8424, RBD=14.0858). Anti-COVID-19 antibody negative at Week 0 is defined separately for spike and RBD. Seroconversion was defined as having a result greater than the positive threshold at the Week 4 visit.
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants who were anti-COVID-19 antibody negative (by either Wu-1 full-length spike or RBD) at Week 0 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 0 | 3 | 4 | 1 | 1 | 3 | 6 | 4 | 38 | 42 | 7
Participants
  Seroconverted, Wu-1 Full-Length Spike: number analyzed (Participants) | 2 | 0 | 2 | 4 | 1 | 1 | 2 | 6 | 4 | 38 | 34 | 7
  Seroconverted, Wu-1 Full-Length Spike | 2 |  | 2 | 3 | 1 | 1 | 2 | 3 | 3 | 13 | 10 | 2
  Seroconverted, Receptor Binding Domain (RBD): number analyzed (Participants) | 2 | 0 | 3 | 4 | 1 | 1 | 3 | 5 | 3 | 38 | 42 | 7
  Seroconverted, Receptor Binding Domain (RBD) | 2 |  | 2 | 3 | 1 | 1 | 3 | 2 | 2 | 12 | 12 | 1

5. Secondary Outcome: Percentage of Stage 2 Adult Participants Who Seroconverted
Description: as for outcome 4
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants who were anti-COVID-19 antibody negative (by Wu-1 full-length spike or RBD) at Week 0 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 41 | 2 | 6
Participants
  Seroconverted, Wu-1 Full-Length Spike: number analyzed (Participants) | 2 | 1 | 0 | 0 | 38 | 2 | 4
  Seroconverted, Wu-1 Full-Length Spike | 1 | 0 |  |  | 7 | 0 | 0
  Seroconverted, Receptor Binding Domain (RBD) | 1 | 1 | 1 |  | 4 | 0 | 0

6. Secondary Outcome: Fold Increase in Stage 1 Adult Anti-COVID-19 Antibody Levels
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center Meso Scale Discovery 3 plex assay. For concentrations below the lower limit of detection (LLOD), numeric values equivalent to LLOD/2 were assigned; concentrations above the upper limit of quantification were reported without adjustments. Antibody results collected after a documented COVID-19 infection, monoclonal antibody use, or a COVID-19 vaccine given off-study were excluded from the analyses. Participants with missing antibody data were considered missing-completely-at-random. Fold increase was assessed in the subgroup of participants who were anti-COVID-19 antibody positive at Week 0; defined as having a result greater than the positive threshold value (spike=10.8424, RBD=14.0858). Anti-COVID-19 antibody positive at Week 0 is defined separately for spike and RBD. Fold increase = (antibody response at Week 4)/(antibody response at Week 0).
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants who were anti-COVID-19 antibody positive (by Wu-1 full-length spike or RBD) at Week 0 were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Change
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 0 | 1 | 6 | 5 | 1 | 2 | 1 | 5 | 7 | 2 | 11 | 1
Fold Change
  Fold Change, Wu-1 Full-Length Spike: number analyzed (Participants) | 0 | 1 | 6 | 5 | 1 | 2 | 1 | 4 | 6 | 2 | 11 | 1
  Fold Change, Wu-1 Full-Length Spike |  | 12.31 (NA) — Sample size didn't support displaying the descriptive statistic | 35.78 (326.98) | 65.38 (165.08) | 3.97 (NA) — Sample size didn't support displaying the descriptive statistic | 66.34 (30.51) | 111.83 (NA) — Sample size didn't support displaying the descriptive statistic | 99.52 (168.72) | 95.54 (75.93) | 2.58 (257.03) | 4.09 (1485.84) | 2.91 (NA) — Sample size didn't support displaying the descriptive statistic
  Fold Change, Receptor Binding Domain (RBD): number analyzed (Participants) | 0 | 1 | 5 | 5 | 1 | 2 | 0 | 5 | 7 | 2 | 3 | 1
  Fold Change, Receptor Binding Domain (RBD) |  | 16.7 (NA) — Sample size didn't support displaying the descriptive statistic | 85.53 (101.49) | 35.32 (358.06) | 9.3 (NA) — Sample size didn't support displaying the descriptive statistic | 85.18 (53.39) |  | 67.9 (142.36) | 80.66 (115.89) | 4.99 (1175.81) | 1.95 (86.7) | 4.48 (NA) — Sample size didn't support displaying the descriptive statistic

7. Secondary Outcome: Fold Increase in Stage 2 Adult Anti-COVID-19 Antibody Levels
Description: as for outcome 6
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Change
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 7 | 4 | 8 | 6 | 13 | 0 | 16
Fold Change
  Fold Change, Wu-1 Full-Length Spike | 54.15 (103.71) | 9.97 (146.18) | 49.62 (603.67) | 5.17 (278.52) | 2.74 (287.75) |  | 0.82 (12.82)
  Fold Change, Receptor Binding Domain (RBD): number analyzed (Participants) | 7 | 3 | 7 | 6 | 10 | 0 | 14
  Fold Change, Receptor Binding Domain (RBD) | 93.53 (111.68) | 17.65 (309.52) | 44.49 (716.62) | 5.46 (299.38) | 4.02 (648.61) |  | 0.8 (10.47)

8. Secondary Outcome: Change in Stage 1 Adult Anti-COVID-19 Antibody Response
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center (NIAID-VRC) Meso Scale Discovery (MSD) 3 plex assay (Wu-1 full-length spike, receptor binding domain (RBD), and N proteins). Wu-1 full-length spike and RBD were used to assess vaccine response. For concentrations below the lower limit of detection (LLOD), numeric values equivalent to LLOD/2 were assigned; concentrations above the upper limit of quantification were reported without adjustments. Antibody results collected after a documented COVID-19 infection, monoclonal antibody use, or a COVID-19 vaccine given off-study were excluded from the analyses. Participants with missing anti-COVID-19 antibody response data were considered to be missing-completely-at-random.
Time Frame: Week 0 and Weeks 4 and 12 Status Post Receipt of COVID-19 Vaccination
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
IU/mL
  Week 0, Wu-1 Full-Length Spike | 2.52 (221.96) | 224.49 (NA) — Sample size didn't support displaying the descriptive statistic | 14.52 (196.41) | 8.67 (1803.07) | 16.83 (279.39) | 18.83 (87.58) | 5.31 (107.14) | 7.22 (121.07) | 11.72 (117.09) | 0.95 (289.7) | 1.99 (1091.74) | 2.25 (1536.33)
  Week 4, Wu-1 Full-Length Spike | 321.14 (10668.22) | 2763.2 (NA) — Sample size didn't support displaying the descriptive statistic | 518.82 (452.03) | 632.72 (2925.17) | 296.41 (70.11) | 1681.23 (20.2) | 1104.81 (436.85) | 459.48 (1333.45) | 2211.08 (252.38) | 4.88 (5181.02) | 8.02 (8352.66) | 9.03 (62605.68)
  Week 12, Wu-1 Full-Length Spike | 356.28 (6108.73) | 3121.73 (NA) — Sample size didn't support displaying the descriptive statistic | 331.49 (333.85) | 626.32 (650.04) | 232.72 (97.53) | 660.98 (91.92) | 296.69 (481.82) | 362.53 (214.09) | 597.3 (216.04) | 6.88 (3896.56) | 6.28 (6838.48) | 5.59 (1429421.94)
  Week 0, Receptor Binding Domain (RBD) | 6.45 (39.72) | 207.45 (NA) — Sample size didn't support displaying the descriptive statistic | 12.34 (142.28) | 12.36 (424.64) | 12.27 (67.11) | 24.54 (92.01) | 6.65 (45.13) | 13.88 (65.76) | 17.42 (119.26) | 2.45 (134.77) | 1.74 (206.49) | 7.53 (282.2)
  Week 4, Receptor Binding Domain (RBD) | 434.06 (157747.37) | 3464.82 (NA) — Sample size didn't support displaying the descriptive statistic | 458.18 (1185.39) | 491.61 (7488.68) | 355.86 (131.08) | 2266.65 (59.16) | 1751.42 (544.5) | 601.12 (797.51) | 3074.6 (246.3) | 8.84 (943.12) | 7.73 (3104.64) | 16.64 (4363.12)
  Week 12, Receptor Binding Domain (RBD) | 466.11 (104511.25) | 3734.51 (NA) — Sample size didn't support displaying the descriptive statistic | 272.17 (920.54) | 617.58 (630.84) | 276.55 (225.66) | 926.48 (162) | 497.09 (542.78) | 456.9 (123.89) | 948.78 (219.75) | 10.36 (989.47) | 6.61 (2278.71) | 12.37 (102810.04)

9. Secondary Outcome: Change in Stage 2 Adult Anti-COVID-19 Antibody Response
Description: as for outcome 8
Time Frame: Week 0 and Weeks 4 and 12 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
IU/mL
  Week 0, Wu-1 Full-Length Spike | 22.14 (1247.32) | 48.64 (23319.38) | 127.11 (3076.50) | 228.43 (163.73) | 3.83 (1803.22) | 0.33 (144.78) | 139.71 (8202.42)
  Week 4, Wu-1 Full-Length Spike | 1329.5 (3501.10) | 306.1 (1263457.31) | 6307.1 (166.16) | 1122.85 (156.9) | 9.67 (7718.35) | 0.33 (145.66) | 137.36 (5885.99)
  Week 12, Wu-1 Full-Length Spike | 684.1 (7400.94) | 205.05 (683623.84) | 1143.73 (109.59) | 701.21 (193.34) | 13.88 (6077.43) | 0.15 (NA) — Sample size didn't support displaying the descriptive statistic | 88.11 (4049.13)
  Week 0, Receptor Binding Domain (RBD) | 18.28 (314.85) | 40.85 (5113.92) | 136.55 (5462.96) | 312.05 (167.64) | 3.87 (933.74) | 1.17 (58.88) | 195.64 (32100.88)
  Week 4, Receptor Binding Domain (RBD) | 1583.14 (2496.89) | 593.17 (173461.30) | 8464.11 (216.65) | 1668.91 (162.22) | 7.56 (4854.01) | 1.24 (69.04) | 187.34 (21600.14)
  Week 12, Receptor Binding Domain (RBD) | 812.4 (6728.02) | 311.56 (120989.28) | 1458.9 (113.83) | 1030.47 (203.85) | 11.4 (3794.97) | 0.8 (NA) — Sample size didn't support displaying the descriptive statistic | 123.87 (9374.45)

10. Secondary Outcome: Fold Inhibition of ACE2 Binding to SARS-CoV-2 Variant Antigens by Stage 1 Adult Samples
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center (NIAID-VRC) Meso Scale Discovery (MSD) V-Plex ACE2 neutralization assay which measure antibodies that block the binding of angiotensin-converting enzyme 2 (ACE2) to the SARS-CoV-2 Spike antigens, including variants of the SARS-CoV-2 virus according to the manufacturer's instruction (MSD Catalog # K15654U). Antibody results collected after a documented COVID-19 infection, monoclonal antibody use, or a COVID-19 vaccine given off-study were excluded from the analyses. Participants with missing anti-COVID-19 antibody response data were considered to be missing-completely-at-random. Results are reported as fold inhibition by a sample relative to signal from a 'diluent only' control (maximum ACE2 binding to antigen). Highly neutralizing samples show high fold inhibition whereas negative or low samples show low fold inhibition of ACE2 binding.
Time Frame: Week 0 and Weeks 4 and 12 Status Post Receipt of COVID-19 Vaccination
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Inhibition
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Fold Inhibition
  Week 0 | 1 (0) | 2 (NA) — Sample size didn't support displaying the descriptive statistic | 1 (0) | 1.08 (23.42) | 1 (0.00) | 1 (0) | 1 (0) | 1 (0) | 1 (0) | 1 (0) | 1.02 (10.36) | 1.09 (24.88)
  Week 4 | 15.03 (154928.64) | 18 (NA) — Sample size didn't support displaying the descriptive statistic | 5.96 (291.28) | 9.49 (577.34) | 3.46 (91.02) | 5.52 (255.65) | 40.15 (914418.24) | 6.16 (383.45) | 24.88 (2444.17) | 1.16 (38.70) | 1.14 (31.58) | 1.31 (73.48)
  Week 12 | 9.11 (13182.95) | 30 (NA) — Sample size didn't support displaying the descriptive statistic | 2.99 (249.41) | 3.56 (135.35) | 4.47 (162.84) | 1.59 (41.68) | 5.67 (9124.55) | 2.16 (63.89) | 4.25 (203.12) | 1.08 (22.87) | 1.55 (653.94) | 1.59 (94.74)

11. Secondary Outcome: Fold Inhibition of ACE2 Binding to SARS-CoV-2 Variant Antigens by Stage 2 Adult Samples
Description: as for outcome 10
Time Frame: Week 0 and Weeks 4 and 12 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Inhibition
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Fold Inhibition
  Week 0 | 1 (0.00) | 1.64 (51.25) | 3.2 (9598.10) | 1.62 (59.19) | 1.14 (86.32) | 1 (0) | 9.42 (412.99)
  Week 4 | 23.32 (651.97) | 15.31 (6552.75) | 109.39 (1119.69) | 7.34 (1124.11) | 1.54 (195.75) | 1 (0) | 6.6 (268.60)
  Week 12 | 7.61 (701.06) | 10.34 (4255.15) | 5.71 (319.78) | 4.03 (451.42) | 1.43 (117.21) | 1 (NA) — Sample size didn't support displaying the descriptive statistic | 2.9 (100.15)

12. Secondary Outcome: Change in Stage 1 Adult Disease Activity as Measured by the Clinical Global Impression of Change (CGI-C)
Description: The Clinical Global Impression of Change (CGI-C) is the clinician's global impression of a participant's clinical condition in terms of change relative to the start of treatment. Change is rated on a 7-point scale from 1 (very much improved) to 7 (very much worse). Higher score = more affected.
Time Frame: Weeks 4 Status Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 1 | 3 | 3 | 9 | 10 | 38 | 44 | 8
Participants
  Very much improved | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Much improved | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Minimally improved | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 0
  No change | 1 | 0 | 7 | 6 | 0 | 3 | 2 | 7 | 7 | 26 | 42 | 8
  Minimally worse | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 6 | 2 | 0
  Much worse | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Change in Stage 2 Adult Disease Activity After Receipt of Additional Doses of COVID-19 Vaccine as Measured by the Clinical Global Impression of Change (CGI-C)
Description: as for outcome 12
Time Frame: Weeks 4 Status Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 5 | 52 | 2 | 20
Participants
  Very much improved | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Much improved | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Minimally improved | 2 | 1 | 0 | 0 | 3 | 0 | 0
  No change | 7 | 3 | 8 | 4 | 44 | 2 | 18
  Minimally worse | 0 | 1 | 0 | 1 | 5 | 0 | 2
  Much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Change in Adult Stage 1 Disease Activity as Measured by the Physician's Global Assessment
Description: The Physician's Global Assessment of the participant's current disease activity is assessed on a 10 cm linear horizontal visual analog scale, where the left hand extreme of the line is considered "Very Good" (0 cm, no disease activity) and the right hand extreme is considered "Very Bad" (10 cm, severe disease activity).
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
cm
  Week 0 | 1.1 (1.3) | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 1.2 (0.9) | 2.5 (2.6) | 1.9 (1.5) | 1.2 (0.6) | 1.2 (1.6) | 1.5 (1.2) | 1.2 (1.8) | 1.1 (1.5) | 1.6 (2.6) | 1.3 (1.8)
  Week 4 | 2.8 (1.6) | 0.4 (NA) — Sample size didn't support displaying the descriptive statistic | 1.6 (1.2) | 1.7 (1.9) | 4.5 (2.8) | 0.7 (0.8) | 0.5 (0.8) | 1.2 (1.2) | 1.3 (1.6) | 1.3 (1.7) | 0.5 (1) | 0.7 (1.1)
  Week 12 | 2.1 (2.7) | 0.2 (NA) — Sample size didn't support displaying the descriptive statistic | 1.6 (1.1) | 1.2 (1.3) | 3.4 (4.4) | 1 (0.7) | 1.8 (0.8) | 0.7 (0.9) | 1.3 (1.1) | 1.6 (1.9) | 0.8 (1.5) | 1.1 (1.8)

15. Secondary Outcome: Change in Adult Stage 2 Disease Activity After Receipt of Additional Doses of COVID-19 Vaccine as Measured by the Physician's Global Assessment
Description: as for outcome 14
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
cm
  Week 0 | 1.7 (1.6) | 2.6 (3.1) | 0.4 (0.4) | 1 (0.8) | 1.4 (2) | 0.8 (0.1) | 1.4 (1.1)
  Week 4 | 1.7 (1.7) | 3.4 (2.4) | 0.6 (0.5) | 0.9 (0.6) | 1.54 (1.8) | 1.1 (0.9) | 1.3 (1.6)
  Week 12 | 1.3 (1.2) | 1.8 (2.1) | 0.5 (0.4) | 1 (0.8) | 1.6 (1.8) | 0.2 (0.1) | 1 (1.4)

16. Secondary Outcome: Change in Disease Activity in Stage 1 Adult Participants With Systemic Lupus Erythematosus (SLE) as Measured by Hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI)
Description: The Hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI) is a validated, physician-based assessment tool used to measure the extent of lupus disease activity within the past 28 days. hSLEDAI total score is a weighted sum of the presence of 24 lupus disease symptoms and ranges from 0 to 105, with higher scores indicating more lupus disease activity present.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants with Systemic Lupus Erythematosus (SLE) are included in the analysis.
Measure: Mean (Standard Deviation); unit: hSLEDAI Score
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1 | 3 | 3 | 2 | 2 | 1
hSLEDAI Score
  Week 0: number analyzed (Participants) | 1 | 1 | 6 | 7 | 1 | 3 | 3 | 2 | 1 | 1
  Week 0 | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 2 (2.19) | 7.83 (6.21) | 4 (NA) — Sample size didn't support displaying the descriptive statistic | 2 (3.46) | 0.67 (1.15) | 2 (2.83) | 4 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4 | 4 (NA) — Sample size didn't support displaying the descriptive statistic | 2 (NA) — Sample size didn't support displaying the descriptive statistic | 3.4 (2.97) | 5.57 (4.31) | 6 (NA) — Sample size didn't support displaying the descriptive statistic | 2.67 (3.06) | 0.67 (1.15) | 3 (4.24) | 4 (2.83) | 2 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12: number analyzed (Participants) | 1 | 1 | 6 | 7 | 1 | 3 | 3 | 1 | 2 | 1
  Week 12 | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 2 (NA) — Sample size didn't support displaying the descriptive statistic | 3.33 (3.27) | 5.57 (6.11) | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (0) | 1.33 (2.31) | 4 (NA) — Sample size didn't support displaying the descriptive statistic | 4 (2.83) | 0 (NA) — Sample size didn't support displaying the descriptive statistic

17. Secondary Outcome: Change in Disease Activity in Stage 2 Adult Participants With Systemic Lupus Erythematosus (SLE) as Measured by Hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI)
Description: as for outcome 16
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hSLEDAI Score
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT)
Number analyzed (Participants) | 3 | 2 | 3
hSLEDAI Score
  Week 0: number analyzed (Participants) | 3 | 1 | 3
  Week 0 | 4 (4) | 2 (NA) — Sample size didn't support displaying the descriptive statistic | 4 (4.4)
  Week 4 | 0.7 (1.2) | 4 (2.8) | 4.3 (4)
  Week 12 | 0.7 (1.2) | 2 (0) | 3 (1.4)

18. Secondary Outcome: Change in Disease Activity in Stage 1 Adult Participants With Systemic Lupus Erythematosus (SLE) as Measured by the Thanou Modified SELENA-SLEDAI Flare Index
Description: The Thanou Modified Safety of Estrogens in Lupus Erythematosus: National Assessment- Hybrid Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) assesses systemic lupus erythematosus (SLE) disease activity and categorizes mild/moderate or severe flares based on changes in the SLEDAI score, the Physician's Global Assessment (PGA), other disease activity criteria, and hospitalization due to SLE. The hSLEDAI is a validated, physician-based assessment tool used to measure the extent of lupus disease activity within the past 28 days. hSLEDAI total score is a weighted sum of the presence of 24 lupus disease symptoms and ranges from 0 to 105, with higher scores indicating more lupus disease activity present.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1 | 3 | 3 | 2 | 2 | 1
Participants
  Severe SELENA-SLEDAI Flare at Week 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Severe SELENA-SLEDAI Flare at Week 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe SELENA-SLEDAI Flare at Week 12 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Change in Disease Activity in Stage 2 Adult Participants With Systemic Lupus Erythematosus (SLE) as Measured by the Thanou Modified SELENA-SLEDAI Flare Index
Description: as for outcome 18
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT)
Number analyzed (Participants) | 3 | 2 | 3
Participants
  Severe SELENA-SLEDAI Flare at Week 0 | 0 | 0 | 0
  Severe SELENA-SLEDAI Flare at Week 4 | 0 | 0 | 0
  Severe SELENA-SLEDAI Flare at Week 12 | 0 | 0 | 0

20. Secondary Outcome: Change in Disease Activity in Stage 1 Adult Participants With Rheumatoid Arthritis (RA) as Measured by Disease Activity Score 28 C-reactive Protein (DAS28-CRP)
Description: The Disease Activity Score 28 C-reactive Protein (DAS28-CRP) is: a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables(the number of tender joints out of 28, the number of swollen joints out of 28 joints, serum C-reactive protein in mg/L (CRP) and subject assessment of disease activity measure on a visual analogue scale (VAS) of 100 mm). Reference: van Gestel AM et al. Arthritis Rheum.1998; 41(10): 1845-50.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants with Rheumatoid Arthritis (RA) are included in the analysis.
Measure: Mean (Standard Deviation); unit: DAS28-CRP Score
Arm/Group | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT)
Number analyzed (Participants) | 3 | 3 | 7 | 7 | 10 | 8
DAS28-CRP Score
  Week 0: number analyzed (Participants) | 3 | 1 | 7 | 7 | 10 | 8
  Week 0 | 2.7 (1.1) | 2.5 (NA) — Sample size didn't support displaying the descriptive statistic | 2.1 (0.8) | 2.7 (1.3) | 3.1 (1.4) | 3.3 (1.5)
  Week 4 | 3 (0.7) | 2.6 (0.9) | 1.6 (0.6) | 2.8 (1.1) | 3.3 (1.3) | 3.3 (1.1)
  Week 12: number analyzed (Participants) | 3 | 1 | 7 | 7 | 10 | 8
  Week 12 | 3.5 (0) | 3.5 (NA) — Sample size didn't support displaying the descriptive statistic | 2.1 (1.1) | 2.8 (1) | 3.4 (2.3) | 3.2 (1.7)

21. Secondary Outcome: Change in Disease Activity in Stage 2 Adult Participants With Rheumatoid Arthritis (RA) as Measured by Disease Activity Score 28 C-reactive Protein (DAS28-CRP)
Description: as for outcome 20
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: DAS28-CRP Score
Arm/Group | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 8 | 6 | 9 | 5
DAS28-CRP Score
  Week 0 | 1.9 (0.6) | 1.8 (0.7) | 2.8 (1.2) | 3 (0.8)
  Week 4 | 2.1 (0.5) | 2 (0.7) | 2.6 (1) | 2.6 (0.9)
  Week 12 | 1.9 (0.4) | 2 (0.8) | 3 (1.2) | 2.3 (0.4)

22. Secondary Outcome: Change in Disease Activity in Stage 1 Adult Participants With Systemic Sclerosis (SSc) as Measured by Disease Flare Activity
Description: Severe disease flare included onset of new or significant worsening of internal organ involvement requiring hospitalization or change in treatment. Internal organ involvement included scleroderma renal crisis, interstitial lung disease, left or right sided heart failure, pulmonary arterial hypertension on right-sided heart catheterization or other worsening of internal organs.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants with Systemic Sclerosis (SSc) are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT)
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 1
Participants
  Severe Flare at Week 0 | 0 | 0 | 0 | 0 | 0
  Severe Flare at Week 4 | 0 | 0 | 0 | 0 | 0
  Severe Flare at Week 12 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Change in Disease Activity in Stage 2 Adult Participants With Systemic Sclerosis (SSc) as Measured by Disease Flare Activity
Description: as for outcome 22
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 6 | 3 | 1
Participants
  Severe Flare at Week 0 | 0 | 0 | 0
  Severe Flare at Week 4 | 0 | 0 | 0
  Severe Flare at Week 12 | 0 | 0 | 0

24. Secondary Outcome: Change in Disease Activity in Stage 1 Adult Participants With Pemphigus as Measured by Disease Area Index (PDAI) for Pemphigus
Description: The Pemphigus Disease Area Index (PDAI) was developed by the International Pemphigus Committee and measures both activity of and damage due to pemphigus on the skin, scalp, and mucous membranes. Total scores can range from 0 to a possible 263 maximum score, with 250 points representing disease activity (120 points for skin activity, 10 points for scalp activity, and 120 points for mucosal activity) and 13 points representing disease damage. Higher scores reflect worse disease.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants with Pemphigus are included in the analysis.
Measure: Mean (Standard Deviation); unit: PDAI Total Activity Score
Arm/Group | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT)
Number analyzed (Participants) | 1 | 2
PDAI Total Activity Score
  Week 0 | 1 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (0)
  Week 4 | 5 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (0)
  Week 12 | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 1 (1.41)

25. Secondary Outcome: Change in Disease Activity in Stage 2 Adult Participants With Pemphigus as Measured by Disease Area Index (PDAI) for Pemphigus
Description: as for outcome 24
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: PDAI Total Activity Score
Arm/Group | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 4 | 2
PDAI Total Activity Score
  Week 0 | 0 (0) | 0 (0)
  Week 4 | 0 (0) | 0 (0)
  Week 12 | 0 (0) | 0 (0)

26. Secondary Outcome: Change in Disease Activity in Stage 1 Adult Participants With Multiple Sclerosis (MS) as Measured by Physician Assessed Relapse for MS
Description: Relapse required: either criteria (a) with investigator determination of relapse or criteria (a) and (b): (a) New, recurrent or worsening neurological symptoms attributable to MS, that meet all of the following: i. Appeared or evolved subacutely (over <3 months). ii. Persisting >24 hours. iii. Can't be attributed to confounding factors. iv. Occur ≥30 days after onset of a prior confirmed relapse. (b) New, recurrent or worsening neurological symptoms accompanied by corresponding objective worsening on neurologic examination with an increase of any one of the following compared to the immediate prior assessment: i. ≥0.5 step(s) on the Expanded Disability Status Scale (EDSS), ii. ≥2 points on one Functional Systems Score (FSS), iii. ≥1 point on two or more FSS. Episodic spasms, sexual dysfunction, fatigue, mood change, or bladder/bowel urgency or incontinence will not suffice to establish relapse. Sexual dysfunction and fatigue will not contribute to the EDSS/FSS for assessing relapse.
Time Frame: Screening and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were randomized or allocated and received study vaccine in the study. Only participants with Multiple Sclerosis (MS) are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 26 | 34 | 7
Participants
  MS Relapse at Screening | 0 | 0 | 0
  MS Relapse at Week 4 | 0 | 0 | 0
  MS Relapse at Week 12 | 0 | 0 | 0

27. Secondary Outcome: Change in Disease Activity in Stage 2 Adult Participants With Multiple Sclerosis (MS) as Measured by Physician Assessed Relapse for MS
Description: as for outcome 26
Time Frame: Screening and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study. Only participants with Multiple Sclerosis (MS) are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 37 | 2 | 12
Participants
  MS Relapse at Screening | 0 | 0 | 0
  MS Relapse at Week 4 | 0 | 0 | 0
  MS Relapse at Week 12 | 0 | 0 | 0

28. Secondary Outcome: Change in Disease Activity in Stage 2 Pediatric Participants With Juvenile Idiopathic Arthritis (JIA) as Measured by the Juvenile Arthritis Disease Activity Score 10 (JADAS10)
Description: The Juvenile Arthritis Disease Activity Score 10-C-reactive Protein (JADAS10-CRP) is a score on a scale (0 to 40) indicating activity of juvenile idiopathic arthritis. Total active joints are scored 0 to 10, with an active joint count >10 scored as 10 points. The Physician's Global Assessment and Patient's Global Assessment are measured on a 0-10 scale (0 cm, no disease activity to 10 cm, worst disease activity). CRP is normalized to a 0 to 10 scale according to the following formula: (CRP (mg/L) - 10)/10. CRP values <10 mg/L are scored as 0, and CRP >110 mg/L are scored as 10. The final score is given by the simple sum of its component. Higher scores indicate worse disease activity.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study. Only participants with Juvenile Idiopathic Arthritis (JIA) are included in the analysis.
Measure: Mean (Standard Deviation); unit: JADAS10 Score
Arm/Group | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1
JADAS10 Score
  Week 0 | 0.8 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4 | 0.6 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12 | 0.4 (NA) — Sample size didn't support displaying the descriptive statistic

29. Secondary Outcome: Change in Adult Stage 1 Disease Activity as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Short Form (Version 2.0) will be used to assess trends over time in this state of health measure. The PROMIS-29 consists of 7 domains related to physical, mental and social health. Raw scores are calculated for each domain and translated into a T-score per the PROMIS-29 scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. Physical Function domain score is presented. A higher score represents better functioning for the Physical Function domain.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
T-Score
  Week 0: number analyzed (Participants) | 1 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
  Week 0 | 37.9 (NA) — Sample size didn't support displaying the descriptive statistic | 43.4 (NA) — Sample size didn't support displaying the descriptive statistic | 47.6 (10.1) | 40.2 (3.9) | 35.6 (3.3) | 50.1 (6.1) | 39.6 (5) | 48.9 (9) | 41.8 (12) | 43.5 (9.5) | 44.2 (9.9) | 43.5 (11.8)
  Week 4 | 39.8 (0.9) | 41.8 (NA) — Sample size didn't support displaying the descriptive statistic | 48.9 (8.7) | 42.7 (10) | 41.9 (2.1) | 46.5 (2.7) | 42.7 (12.3) | 47.2 (10.5) | 41.7 (10.5) | 43.5 (9.1) | 44.7 (10.5) | 43.6 (11.7)
  Week 12 | 37.3 (0.8) | 56.9 (NA) — Sample size didn't support displaying the descriptive statistic | 47.6 (10.1) | 42.1 (7.7) | 35 (2.4) | 45.3 (0) | 39.3 (7.5) | 46.1 (11.5) | 41.1 (11.9) | 43.5 (9.4) | 44.7 (9.5) | 44.1 (11.9)

30. Secondary Outcome: Change in Adult Stage 2 Disease Activity as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 29
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
T-Score
  Week 0 | 44.9 (7.9) | 46.3 (7.6) | 48.3 (10.4) | 48.3 (8.4) | 45.9 (9.9) | 56.9 (0) | 47.1 (9.5)
  Week 4 | 46.4 (8.5) | 42.5 (10.5) | 48.4 (10.4) | 47.2 (9.4) | 44.9 (9.6) | 56.9 (0) | 48.6 (9.6)
  Week 12 | 45.5 (9.3) | 46.8 (9.3) | 47.6 (9) | 44.2 (8.5) | 43.9 (10) | 51.1 (8.2) | 48.3 (9.4)

31. Secondary Outcome: Change in Adult Stage 1 Disease Activity as Measured by the Patient Global Assessment
Description: The Patient Global Assessment of the participant's current disease activity is assessed on a 10 cm linear horizontal visual analog scale, where the left hand extreme of the line is considered "Very Good" (0 cm, no disease activity) and the right hand extreme is considered "Very Bad" (10 cm, severe disease activity).
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
cm
  Week 0 | 7.2 (2.1) | 3 (NA) — Sample size didn't support displaying the descriptive statistic | 3.1 (2.9) | 3.8 (2.9) | 5.8 (1.8) | 4.8 (1.9) | 5.4 (1.6) | 3.7 (2.4) | 5.1 (3.6) | 3.8 (2.4) | 3.2 (2.9) | 3.9 (3.2)
  Week 4 | 7.9 (0.5) | 6.5 (NA) — Sample size didn't support displaying the descriptive statistic | 2.7 (2.3) | 3.1 (2.3) | 4.9 (4.4) | 6.5 (0.9) | 5.6 (1.8) | 3.6 (2.9) | 4.9 (3.6) | 3.3 (2.6) | 2.6 (2.4) | 3 (2.6)
  Week 12 | 5.8 (1.1) | 7.5 (NA) — Sample size didn't support displaying the descriptive statistic | 3.5 (2.9) | 3.7 (3.2) | 6.2 (1.1) | 4.6 (1.1) | 6.8 (1.5) | 4.3 (3.1) | 4.9 (3) | 3.5 (2.5) | 2.3 (2.2) | 2.3 (2.3)

32. Secondary Outcome: Change in Adult Stage 2 Disease Activity as Measured by the Patient Global Assessment
Description: as for outcome 31
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
cm
  Week 0 | 3.2 (2.6) | 2.7 (3.4) | 3.2 (2.1) | 2.8 (2.6) | 2.7 (2.5) | 2.6 (3.4) | 2.6 (2.6)
  Week 4 | 3 (2.1) | 2.9 (3.1) | 3 (2.5) | 3 (2) | 3 (2.5) | 1 (1.4) | 2.7 (2.9)
  Week 12 | 2.9 (2.7) | 1.8 (2.2) | 3.1 (2.3) | 3.9 (2.7) | 3.1 (2.5) | 2.5 (3.5) | 1.9 (2.2)

33. Secondary Outcome: Change in Stage 1 Adult Disease Activity as Measured by the Patient Global Impression of Change (PGI-C)
Description: The Patient Global Impression of Change (PGI-C) is the participant's global impression of their clinical condition in terms of change relative to the start of treatment. Change is rated on a 7-point scale from 1 (very much improved) to 7 (very much worse). Higher score = more affected.
Time Frame: Weeks 4 Status Post Receipt of COVID-19 Vaccine Dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 9 | 10 | 38 | 44 | 8
Participants
  Very much improved | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Much improved | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Minimally improved | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  No change | 1 | 1 | 8 | 7 | 1 | 2 | 2 | 8 | 6 | 31 | 41 | 7
  Minimally worse | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 5 | 1 | 0
  Much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

34. Secondary Outcome: Change in Stage 2 Adult Disease Activity as Measured by the Patient Global Impression of Change (PGI-C)
Description: as for outcome 33
Time Frame: Weeks 4 Status Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 5 | 52 | 2 | 20
Participants
  Very much improved | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Much improved | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Minimally improved | 2 | 2 | 1 | 0 | 3 | 0 | 0
  No change | 7 | 2 | 7 | 5 | 46 | 2 | 19
  Minimally worse | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Much worse | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Very much worse | 0 | 1 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Percent of Stage 1 Adult Participants Who Experience Any Grade 1 or Higher Adverse Events Related to Study Vaccine
Description: All unsolicited adverse events (AEs) (all grades) were collected from Day 1 through Day 28; solicited AEs were collected if they were ongoing at Day 7 (post vaccination); any flares of a secondary autoimmune disease, serious AEs, medically attended AEs, new onset chronic medical conditions, and COVID-19 infections were collected from Day 1 through the end of the participant's study participation. All AEs were classified by system organ class (SOC) and preferred term, according to a standardized thesaurus (Medical Dictionary for Regulatory Activities [MedDRA] version 24.0. Related AEs were defined as "possibly related" (the AE has a reasonable possibility to be related; there is evidence to suggest a causal relationship) or "related" (the adverse event is clearly related). Severity was assessed according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Time Frame: Up to Week 48 post study vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0

36. Secondary Outcome: Percent of Stage 2 Adult Participants Who Experience Any Grade 1 or Higher Adverse Events Related to Study Vaccine
Description: as for outcome 35
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Participants | 2 | 0 | 1 | 1 | 4 | 0 | 0

37. Secondary Outcome: Percent of Stage 1 Adult Participants Who Experience Any Serious Adverse Events (SAEs)
Description: An event is considered "serious" if, in the view of either the investigator or Sponsor, it results in any of the following: 1. Death. 2. Life-threatening event: considered "life-threatening" if, in the view of either the investigator or Sponsor, its occurrence places the participant at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death. 3. Inpatient hospitalization or prolongation of existing hospitalization. 4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions. 5. Congenital anomaly or birth defect. 6. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Week 48 post study vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 4 | 0

38. Secondary Outcome: Percent of Stage 2 Adult Participants Who Experience Any Serious Adverse Events (SAEs)
Description: as for outcome 37
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Participants | 1 | 1 | 0 | 0 | 6 | 0 | 1

39. Secondary Outcome: Percent of Stage 1 Adult Participants Who Experience Any Medically Attended Adverse Events (MAAEs)
Description: Medically attended adverse event (MAAE) is defined as a hospitalization, emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason that is considered possibly related or related to study vaccine.
Time Frame: Up to Week 48 post study vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

40. Secondary Outcome: Percent of Stage 2 Adult Participants Who Experience Any Medically Attended Adverse Events (MAAEs)
Description: as for outcome 39
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Percent of Stage 1 Adult Participants Who Experience Any New Onset Chronic Medical Conditions (NOCMCs)
Description: A new onset chronic medical condition (NOCMC) is defined as any new ICD diagnosis (per current International Statistical Classification of Diseases and Related Health Problems) that is applied to the study participant during the course of the study, after receipt of the vaccine, that is expected to continue for at least 3 months and requires continued health care intervention.
Time Frame: Up to Week 48 post study vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0

42. Secondary Outcome: Percent of Stage 2 Adult Participants Who Experience Any New Onset Chronic Medical Conditions (NOCMCs)
Description: as for outcome 41
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Participants | 0 | 0 | 0 | 0 | 2 | 0 | 1

43. Secondary Outcome: Percent of Stage 1 Adult Participants Who Experience Any Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Infection
Description: Efficacy measure.
Time Frame: Up to Week 48 post study vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT)
Number analyzed (Participants) | 2 | 1 | 8 | 9 | 2 | 3 | 3 | 10 | 10 | 40 | 45 | 8
Participants | 1 | 0 | 3 | 3 | 0 | 1 | 0 | 3 | 6 | 14 | 12 | 6

44. Secondary Outcome: Percent of Stage 2 Adult Participants Who Experience Any Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Infection
Description: COVID-19 infections (all grades) were confirmed by molecular COVID-19 testing. AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 24.0.
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT)
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 53 | 2 | 20
Participants | 2 | 1 | 1 | 3 | 20 | 0 | 6

45. Secondary Outcome: Percentage of Stage 2 Pediatric Participants Who Seroconverted
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center Meso Scale Discovery 3 plex assay. For concentrations below the lower limit of detection (LLOD), numeric values equivalent to LLOD/2 were assigned; concentrations above the upper limit of quantification were reported without adjustments. Antibody results collected after a documented COVID-19 infection, monoclonal antibody use, or a COVID-19 vaccine given off-study were excluded from the analyses. Participants with missing antibody data were considered missing-completely-at-random. Seroconversion was assessed in the subgroup of participants who were anti-COVID-19 antibody negative at Week 0; defined as a result less than or equal to the positive threshold value (spike=10.8424, RBD=14.0858), defined independently for spike and RBD. Seroconversion was defined as having a result greater than the positive threshold at the Week 4 visit.
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study. Only participants who were anti-COVID-19 antibody negative at Week 0 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA)
Number analyzed (Participants) | 1
Participants | 0

46. Secondary Outcome: Fold Increase in Stage 2 Pediatric Anti-COVID-19 Antibody Levels
Description: Antibody response was measured using the National Institute of Allergy and Infectious Disease Vaccine Research Center Meso Scale Discovery 3 plex assay. For concentrations below the lower limit of detection (LLOD), numeric values equivalent to LLOD/2 were assigned; concentrations above the upper limit of quantification were reported without adjustments. Antibody results collected after a documented COVID-19 infection, monoclonal antibody use, or a COVID-19 vaccine given off-study were excluded from the analyses. Participants with missing antibody data were considered missing-completely-at-random. Fold increase was assessed in the subgroup of participants who were anti-COVID-19 antibody positive at Week 0; defined as having a result greater than the positive threshold value (spike=10.8424, RBD=14.0858), defined independently for spike and RBD. Fold increase = (antibody response at Week 4)/(antibody response at Week 0).
Time Frame: Week 4 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study. Only participants who were anti-COVID-19 antibody positive at Week 0 were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Change
Arm/Group | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1
Fold Change
  Fold Change, Wu-1 Full-Length Spike | 149.84 (NA) — Sample size didn't support displaying the descriptive statistic
  Fold Change, Receptor Binding Domain (RBD) | 112.05 (NA) — Sample size didn't support displaying the descriptive statistic

47. Secondary Outcome: Change in Stage 2 Pediatric Anti-COVID-19 Antibody Response
Description: as for outcome 8
Time Frame: Week 0 and Weeks 4 and 12 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
IU/mL
  Week 0, Wu-1 Full-Length Spike | 1.27 (NA) — Sample size didn't support displaying the descriptive statistic | 123.28 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4, Wu-1 Full-Length Spike | 6.53 (NA) — Sample size didn't support displaying the descriptive statistic | 18473.06 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12, Wu-1 Full-Length Spike: number analyzed (Participants) | 0 | 1
  Week 12, Wu-1 Full-Length Spike |  | 3583.89 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 0, Receptor Binding Domain (RBD) | 2.49 (NA) — Sample size didn't support displaying the descriptive statistic | 175.7 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4, Receptor Binding Domain (RBD) | 10.65 (NA) — Sample size didn't support displaying the descriptive statistic | 19688.14 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12, Receptor Binding Domain (RBD): number analyzed (Participants) | 0 | 1
  Week 12, Receptor Binding Domain (RBD) |  | 3664.63 (NA) — Sample size didn't support displaying the descriptive statistic

48. Secondary Outcome: Fold Inhibition of ACE2 Binding to SARS-CoV-2 Variant Antigens by Stage 2 Pediatric Samples
Description: as for outcome 10
Time Frame: Week 0 and Weeks 4 and 12 Status Post Receipt of COVID-19 Vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Inhibition
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Fold Inhibition
  Week 0 | 1 (NA) — Sample size didn't support displaying the descriptive statistic | 1 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4 | 1 (NA) — Sample size didn't support displaying the descriptive statistic | 722 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12: number analyzed (Participants) | 0 | 1
  Week 12 |  | 158 (NA) — Sample size didn't support displaying the descriptive statistic

49. Secondary Outcome: Change in Stage 2 Pediatric Disease Activity After Receipt of Additional Doses of COVID-19 Vaccine as Measured by the Clinical Global Impression of Change (CGI-C)
Description: as for outcome 12
Time Frame: Weeks 4 Status Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants
  Very much improved | 0 | 0
  Much improved | 0 | 0
  Minimally improved | 0 | 0
  No change | 1 | 0
  Minimally worse | 0 | 1
  Much worse | 0 | 0
  Very much worse | 0 | 0

50. Secondary Outcome: Change in Pediatric Stage 2 Disease Activity After Receipt of Additional Doses of COVID-19 Vaccine as Measured by the Physician's Global Assessment
Description: as for outcome 14
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
cm
  Week 0 | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 0.8 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4 | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 0.6 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12 | 0 (NA) — Sample size didn't support displaying the descriptive statistic | 0.4 (NA) — Sample size didn't support displaying the descriptive statistic

51. Secondary Outcome: Change in Disease Activity in Stage 2 Pediatric Participants With Systemic Lupus Erythematosus (SLE) as Measured by Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K
Description: The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K is a validated, physician-based assessment tool used to measure the extent of lupus disease activity within the past 28 days. SLEDAI-2K total score is a weighted sum of the presence of 24 lupus disease symptoms and ranges from 0 to 105, with higher scores indicating more lupus disease activity present.
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study. Only participants with Systemic Lupus Erythematosus (SLE) are included in the analysis.
Measure: Mean (Standard Deviation); unit: SLEDAI-2K Score
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA)
Number analyzed (Participants) | 1
SLEDAI-2K Score
  Week 0 | 2 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4 | 2 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12 | 0 (NA) — Sample size didn't support displaying the descriptive statistic

52. Secondary Outcome: Change in Pediatric Stage 2 Disease Activity as Measured by the Patient Global Assessment
Description: as for outcome 31
Time Frame: Baseline and Weeks 4, 12 Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
cm
  Week 0 | 5 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 4 | 5 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (NA) — Sample size didn't support displaying the descriptive statistic
  Week 12 | 5 (NA) — Sample size didn't support displaying the descriptive statistic | 0 (NA) — Sample size didn't support displaying the descriptive statistic

53. Secondary Outcome: Change in Stage 2 Pediatric Disease Activity as Measured by the Patient Global Impression of Change (PGI-C)
Description: as for outcome 33
Time Frame: Weeks 4 Status Post Receipt of COVID-19 Vaccine Dose
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants
  Very much improved | 0 | 0
  Much improved | 0 | 0
  Minimally improved | 0 | 0
  No change | 1 | 1
  Minimally worse | 0 | 0
  Much worse | 0 | 0
  Very much worse | 0 | 0

54. Secondary Outcome: Percent of Stage 2 Pediatric Participants Who Experience Any Grade 1 or Higher Adverse Events Related to Study Vaccine
Description: as for outcome 35
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

55. Secondary Outcome: Percent of Stage 2 Pediatric Participants Who Experience Any Serious Adverse Events (SAEs)
Description: as for outcome 37
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

56. Secondary Outcome: Percent of Stage 2 Pediatric Participants Who Experience Any Medically Attended Adverse Events (MAAEs)
Description: as for outcome 39
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

57. Secondary Outcome: Percent of Stage 2 Pediatric Participants Who Experience Any New Onset Chronic Medical Conditions (NOCMCs)
Description: as for outcome 41
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

58. Secondary Outcome: Percent of Stage 2 Pediatric Participants Who Experience Any Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Infection
Description: as for outcome 44
Time Frame: Up to Week 48 post study vaccination
Population: The vaccinated population includes all participants who were allocated and received study vaccine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All unsolicited adverse events (AEs) (all grades) were collected from Day 1 through Day 28; solicited AEs were collected if they were ongoing at Day 7 (post vaccination); any flares of a secondary autoimmune disease, serious AEs, medically attended AEs, new onset chronic medical conditions, and COVID-19 infections were collected from Day 1 through the end of the participant's study participation (up to Week 48).
Description: Adverse events are reported in the vaccinated population, which includes all participants who were randomized or allocated and received study vaccine in the trial. No participants in the "Cohort F, Arm F1: Janssen + Withhold IS (BCDT)" arm were vaccinated.
Groups:
- Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA): Stage 2 adult participants who previously received an mRNA vaccine and who are taking mycophenolate mofetil (MMF) or mycophenolic acid (MPA) (without additional B cell depleting medications or methotrexate) for management of their underlying autoimmune disease, will withhold their cohort-defining immunosuppressive medications (IS) 3 days before and 10 days after receiving a dose of an alternative COVID-19 vaccine (Moderna mRNA-1273 or Pfizer-BioNTech (BNT162b2), per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX): Stage 2 adult participants who previously received an mRNA vaccine and who are taking methotrexate (MTX) (without additional B cell depleting medications or mycophenolate mofetil or mycophenolic acid) for management of their underlying autoimmune disease will withhold their cohort-defining immunosuppressive medications (IS) for at least 7 days before and at least 7 days after receiving a dose of an alternative COVID-19 vaccine (Moderna mRNA-1273 or Pfizer-BioNTech (BNT162b2), but not for more than 21 days total, per protocol instruction. Participants taking additional IS medications (such as tumor necrosis factor [TNF] inhibitors, JAK inhibitors, abatacept, belimumab, etc.) will be required to continue them during the time of the additional vaccine dose.
- Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT): Stage 2 adult participants who previously received an mRNA COVID-19 vaccine and who are taking B cell depletion therapy (BCDT) for management of their underlying autoimmune disease, regardless of whether they are also taking methotrexate (MTX), mycophenolate mofetil (MMF) or mycophenolic acid (MPA), will continue to take their prescribed, cohort-defining, immunosuppressive medications (IS) without alterations in schedule and dosing. Participants who are taking MMF, MPA, or MTX in addition to BCDTs will withhold these medications (MMF, MPA, or MTX) before and after receiving a dose of the alternative COVID-19 vaccine (Moderna mRNA-1273 or Pfizer-BioNTech (BNT162b2), per protocol instruction. MMF and MPA: hold 3 days before and 10 days after vaccine. MTX: hold for at least 7 days before and at least 7 days after vaccine, but not for more than 21 days total.
Arm/Group | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/8 | 0/9 | 0/2 | 0/3 | 0/3 | 0/10 | 0/10 | 0/40 | 0/45 | 0/8 | 0/9 | 0/5 | 0/8 | 0/6 | 0/53 | 0/2 | 0/20 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/8 | 0/9 | 1/2 | 0/3 | 0/3 | 0/10 | 1/10 | 5/40 | 4/45 | 0/8 | 1/9 | 1/5 | 0/8 | 0/6 | 6/53 | 0/2 | 1/20 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 3/8 | 4/9 | 0/2 | 2/3 | 0/3 | 3/10 | 5/10 | 15/40 | 12/45 | 6/8 | 5/9 | 2/5 | 3/8 | 4/6 | 20/53 | 0/2 | 9/20 | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) (N=2) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) (N=1) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) (N=8) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) (N=9) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) (N=2) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) (N=3) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) (N=3) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) (N=10) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) (N=10) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) (N=40) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) (N=45) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) (N=8) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) (N=9) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) (N=5) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) (N=8) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) (N=6) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) (N=53) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) (N=2) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) (N=20) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) (N=1) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX) (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy alcoholic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uhthoff's phenomenon (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A, Arm A1: Moderna mRNA-1273 + Continue IS (MMF or MPA) (N=2) | Cohort A, Arm A4: Moderna mRNA-1273 + Withhold IS (MMF or MPA) (N=1) | Cohort A, Arm A2: Pfizer-BioNTech + Continue IS (MMF or MPA) (N=8) | Cohort A, Arm A5: Pfizer-BioNTech + Withhold IS (MMF or MPA) (N=9) | Cohort A, Arm A6: Janssen + Withhold IS (MMF or MPA) (N=2) | Cohort B, Arm B1: Moderna mRNA-1273 + Continue IS (MTX) (N=3) | Cohort B, Arm B4: Moderna mRNA-1273 + Withhold IS (MTX) (N=3) | Cohort B, Arm B2: Pfizer-BioNTech + Continue IS (MTX) (N=10) | Cohort B, Arm B5: Pfizer-BioNTech + Withhold IS (MTX) (N=10) | Cohort C, Arm C1: Moderna mRNA-1273 + Continue IS (BCDT) (N=40) | Cohort C, Arm C2: Pfizer-BioNTech + Continue IS (BCDT) (N=45) | Cohort C, Arm C3: Janssen + Continue IS (BCDT) (N=8) | Cohort D, Arm D2: Alternative mRNA + Withhold IS (MMF or MPA) (N=9) | Cohort D, Arm D4: Sanofi-GSK + Withhold IS (MMF or MPA) (N=5) | Cohort E, Arm E2: Alternative mRNA + Withhold IS (MTX) (N=8) | Cohort E, Arm E4: Sanofi-GSK + Withhold IS (MTX) (N=6) | Cohort F, Arm F2: Alternative mRNA + Withhold IS (BCDT) (N=53) | Cohort F, Arm F3: Moderna mRNA-1273 + Withhold IS (BCDT) (N=2) | Cohort F, Arm F4: Sanofi-GSK + Withhold IS (BCDT) (N=20) | Cohort D, Arm D2P: Moderna mRNA-1273 + Withhold IS (MMF/MPA) (N=1) | Cohort E, Arm E2P: Moderna mRNA-1273 + Withhold IS (MTX) (N=1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 5 (5) | 14 (15) | 11 (12) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 20 (22) | 0 (0) | 6 (7) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was closed prior to fully enrolling because of slow enrollment due to increasing infections in the general population with resulting elevated antibody titers, changing CDC vaccination recommendations, and vaccine hesitancy. Original enrollment goals were 60 participants per arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT05000216/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT05000216/SAP_002.pdf
  • Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT05000216/ICF_000.pdf